116194 [DTPA-IPV (INFANRIX-IPV)-061] Statistical Analysis Plan Amendment 2 Final

| | Statistical Analysis Flan Amenument 2 Find |
|---|---|
| <b>gsk</b> GlaxoSmithKline | Statistical Analysis Plan |
| Detailed Title: | A phase III, open-label study to assess the immunogenicity and reactogenicity of GSK Biologicals' DTPa-IPV/Hib vaccine administered as a three-dose primary vaccination course at 3, 4.5 and 6 months of age and a booster dose at 18 months of age in healthy infants in Russia. |
| eTrack study number and<br>Abbreviated Title | 116194 [DTPA-IPV (INFANRIX-IPV)-061] |
| Scope: | All analyses as planned per protocol and for study report. |
| Date of Statistical Analysis<br>Plan | First version: 16-Feb-2015 Amendment 1: 10-Aug-2017 Amendment 2: 14-Dec-2017 |
| Co-ordinating author: | PPD (Lead Statistician) and PPD |
| Ç | (Statistician) |
| Reviewed by: | R&D Project Leader) PPD , Clinical Research and Development Lead (CRDL) PPD (peer reviewer statistician) PPD (public disclosure) PPD (Lead statistical analyst) PPD (Global Regulatory Affairs) PPD (Safety Physician) |
| Approved by: | R&D Project Leader) PPD , Clinical Research and Development Lead (CRDL) PPD (Lead Statistician) PPD (Lead statistical analyst) PPD (Scientific writer) |

APP 9000058193 Statistical Analysis Plan Template (Effective date: 14April 2017)

14-DEC-2017 Page 1 of 51

116194 [DTPA-IPV (INFANRIX-IPV)-061] Statistical Analysis Plan Amendment 2 Final

# **TABLE OF CONTENTS**

| | | | | PAGE |
|---|---|---|---|---|
| LIS | T OF A | BBREVI | ATIONS | 7 |
| 1. | DOCU | JMENT H | IISTORY | 9 |
| 2. | CTLIC | V DECIO | iN | 10 |
| ۷. | STUL | DESIG | JN | 10 |
| 3. | OBJE | | | |
| | 3.1. | Primary | objectives | 12 |
| | 3.2. | Second | ary objectives | 12 |
| 4. | ENDF | POINTS | | 12 |
| | 4.1. | Primary | endpoints | 12 |
| | 4.2. | | ary | |
| 5. | ANAL | YSIS SE | TS | 13 |
| | 5.1. | | on | |
| | | 5.1.1. | Total vaccinated cohort (TVC) | |
| | | 5.1.2. | According-to-protocol cohort for analysis of | |
| | | | immunogenicity of the primary epoch | 14 |
| | | 5.1.3. | Total vaccinated cohort for the booster epoch | 14 |
| | | 5.1.4. | According-to-protocol cohort for analysis of | |
| | | | immunogenicity of the booster epoch | 14 |
| | | 5.1.5. | Adapted ATP cohort | 14 |
| | 5.2. | Criteria | for eliminating data from Analysis Sets | |
| | | 5.2.1. | Elimination from Total vaccinated cohort (TVC) | 15 |
| | | 5.2.2. | Elimination from ATP cohort for immunogenicity | 15 |
| | | | 5.2.2.1. Excluded subjects | |
| | | | 5.2.2.2. Right censored Data | 16 |
| | | | 5.2.2.3. Visit-specific censored Data | 17 |
| | 5.3. | Importa | nt protocol deviation not leading to elimination from ATP | |
| | | cohort f | or immunogenicity | 17 |
| 6. | STAT | ISTICAL | ANALYSES | 17 |
| ٥. | 6.1. | | raphy | |
| | 0.1. | 6.1.1. | Analysis of demographics/baseline characteristics planned | |
| | | 0.1.1. | in the protocol | |
| | | 6.1.2. | Additional considerations | |
| | 6.2. | | re | |
| | 0.2. | 6.2.1. | Analysis of exposure planned in the protocol | |
| | | 6.2.2. | Additional considerations | |
| | 6.3. | - | ogenicity | |
| | 0.0. | 6.3.1. | Analysis of immunogenicity planned in the protocol | |
| | | 6.3.2. | Additional considerations | |
| | 6.4. | | s of safety | |
| | | 6.4.1. | Analysis of safety planned in the protocol | |
| | | 6.4.2. | Additional considerations | |
| 7 | ΑΝΔΙ | YSIS INT | FRPRETATION | 21 |

116194 [DTPA-IPV (INFANRIX-IPV)-061] Statistical Analysis Plan Amendment 2 Final

| | Statistical Analysis Plan Americ | ment z rinai |
|---|---|---|
| 8. | CONDUCT OF ANALYSES | |
| | 8.1. Sequence of analyses | 21 |
| | 8.2. Statistical considerations for interim analyses | <mark>22</mark> |
| | 8.3. Statistical considerations for interim analyses | |
| 9. | CHANGES FROM PLANNED ANALYSES | 22 |
| 10. | LIST OF FINAL REPORT TABLES, LISTINGS AND FIGURES | 22 |
| 11. | ANNEX 1 STANDARD DATA DERIVATION RULE AND STATISTICAL | 00 |
| | METHODS | |
| | 11.1. Statistical Method References | |
| | 11.2. Standard data derivation | |
| | 11.2.1. Date derivation | <mark>23</mark> |
| | 11.2.2. Dose number | 24 |
| | 11.2.3. Demography | 24 |
| | 11.2.4. Immunogenicity | |
| | 11.2.5. Safety | |
| 12. | ANNEX 2: SUMMARY ON ELIMINATION CODES | 29 |
| 13 | ANNEX 3: STUDY SPECIFIC MOCK TFL | 29 |

116194 [DTPA-IPV (INFANRIX-IPV)-061] Statistical Analysis Plan Amendment 2 Final

# **LIST OF TABLES**

| | | PAGE |
|---|---|---|
| Table 1 | Study group and epochs foreseen in the study | 11 |
| Table 2 | Study group and treatment foreseen in the study | 11 |
| Table 3 | Blinding of study epochs | 11 |
| Table 4 | Intensity scales to be used by the parent(s)/LAR(s) for solicited symptoms during the solicited follow-up period | 27 |

116194 [DTPA-IPV (INFANRIX-IPV)-061] Statistical Analysis Plan Amendment 2 Final

# **LIST OF TEMPLATES**

| | | PAGE |
|---|---|---|
| Template 1 | Number of subjects enrolled by center – TVC | 30 |
| Template 2 | Number of subjects vaccinated, completed and withdrawn with reason for withdrawal at Visit 3 - TVC | 30 |
| Template 3 | Number of subjects at each visit and list of withdrawn subjects (TVC) | 31 |
| Template 4 | Number of subjects enrolled into the study as well as the number of subjects excluded from ATP analyses with reasons for exclusion | 32 |
| Template 5 | Deviations from specifications for age and intervals between study visits - TVC | 33 |
| Template 6 | Summary of demographic characteristics (ATP cohort for Immunogenicity) | 34 |
| Template 7 | Study population (TVC) | 35 |
| Template 8 | Anti-rotavirus IgA antibody GMC and seropositivity rates – ATP cohort for Immunogenicity | 35 |
| Template 9 | Reverse cumulative distribution curve for anti-rotavirus IgA antibody concentrations at Visit 3 - ATP cohort for Immunogenicity | 36 |
| Template 10 | Number and percentage of subjects who received study vaccine doses - TVC | 37 |
| Template 11 | Compliance in returning symptom sheets - TVC | 37 |
| Template 12 | Incidence and nature of grade 3 symptoms (solicited and unsolicited) reported during the 4-day (Days 0-3) period after vaccination following each dose and overall (Total vaccinated cohort) | 38 |
| Template 13 | Incidence of solicited local symptoms reported during the 4-day (Days 0-3) period after vaccination following each dose and overall (Total vaccinated cohort) | 39 |
| Template 14 | Percentage of doses with solicited general symptom including those rated grade 3 in intensity and those assessed as related to vaccination during the 8-day (Day 1 to Day 8) follow-up period, for each dose in the pooled HRV vaccine liquid formulation group and the HRV vaccine HRV Lyophilised formulation group - TVC | 40 |

116194 [DTPA-IPV (INFANRIX-IPV)-061] Statistical Analysis Plan Amendment 2 Final

| Template 15 | Percentage of subjects reporting each solicited general symptom including those rated grade 3 in intensity and those assessed as related to vaccination during the 8-day (Day 0 to Day 7) follow-up period, for each dose in the pooled HRV vaccine liquid formulation group and the HRV vaccine HRV Lyophilised formulation group - TVC | 41 |
|---|---|---|
| Template 16 | Incidence of any large injection site reaction (defined as a swelling with a diameter > 100 mm, noticeable diffuse swelling or noticeable increase in limb circumference) with onset within 4 days (Day 0–3) after booster vaccination (Total Vaccinated Cohort at Year 9) | 42 |
| Template 17 | Percentage of subjects with grade 3 unsolicited symptoms classified by MedDRA SOC and PT from Day 0 to Day 30 after any vaccination in each HRV vaccine liquid formulation group - TVC. | 43 |
| Template 18 | Percentage of doses with grade 3 unsolicited symptoms classified by MedDRA SOC and PT from Day 0 to Day 30 after vaccination in each HRV vaccine liquid formulation group - TVC | 45 |
| Template 19 | Number (%) of subjects with serious adverse events from first study vaccination up to Visit 3 including number of events reported (TVC) | 46 |
| Template 20 | Subjects with Serious Adverse Events reported up to Visit 3 - TVC | 47 |
| Template 21 | Number and percentage of doses and of subjects who took at least one concomitant medication from Day 0 to Day 7 after vaccination by type in each HRV vaccine liquid formulation group - TVC | 49 |
| Template 22 | Solicited and Unsolicited symptoms experienced by at least 5 % of subjects classified by MedDRA Primary System Organ Class and Preferred Term within the 31-day (Days 0-30) post-vaccination period - AE below 5 % and SAE excluded (Total vaccinated cohort) | 50 |
| Template 23 | Minimum and maximum activity dates (TVC) | 50 |
| Template 24 | Number of enrolled subjects by age category (TVC) | 50 |
| Template 25 | Number of subjects by country | 51 |
| Template 26 | Listing of dropouts due to AEs, SAEs and solicited symptoms (Total cohort) | 51 |

116194 [DTPA-IPV (INFANRIX-IPV)-061] Statistical Analysis Plan Amendment 2 Final

#### LIST OF ABBREVIATIONS

AE Adverse event

ANOVA Analysis of Variance

ATP Per Protocol Set

CI Confidence Interval

CRF Case Report Form

CTRS Clinical Trial Registry Summary

EL.U/ml ELISA unit per milliliter

Eli Type Internal GSK database code for type of elimination code

ELISA Enzyme-linked immunosorbent assay

ES TVC

GE Gastroenteritis

GSK GlaxoSmithKline

iDMC Independent Data Monitoring Committee

IU/ml International units per milliliter

LL Lower Limit of the confidence interval

MedDRA Medical Dictionary for Regulatory Activities

N.A. Not Applicable

PD Protocol Deviation

RV RotaVirus

SAE Serious adverse event

SAP Statistical Analysis Plan

SAS Statistical Analysis Software

SBIR GSK Biological's Internet Randomization System

SD Standard Deviation

116194 [DTPA-IPV (INFANRIX-IPV)-061] Statistical Analysis Plan Amendment 2 Final

SR Study Report

TFL Tables Figures and Listings

TOC Table of Content

UL Upper Limit of the confidence interval

116194 [DTPA-IPV (INFANRIX-IPV)-061] Statistical Analysis Plan Amendment 2 Final

# 1. DOCUMENT HISTORY

| Date | Description | Protocol Version |
|-------------|---------------|------------------------|
| 16-FEB-2015 | first version | Protocol 24-March-2014 |
| 10-AUG-2017 | Amendment 1 | Protocol Amendment 1 |
| | | dated 11 October 2016 |
| 14-DEC-2017 | Amendment 2 | Protocol Amendment 1 |
| | | dated 11 October 2016 |

The SAP amendment 1 was prepared in order to

- Account for the new assay cut-off: During the course of the study, the assays used to measure the anti-D, -T, -PT, -FHA and -PRN IgG concentrations were re-developed and re-validated and both assay units and assay cut-offs were adapted. The new ELISAs for PT, FHA and PRN were calibrated against the WHO International Standard (NIBSC 06/140). This allowed the expression of concentrations measured with the new ELISAs in international units per milliliter (IU/mL) instead of the formerly used ELISA units per milliliter (ELU/mL). The newly validated DTPa ELISA's have a lower assay cut-off as compared to the one described in the protocol. The current assay cut-off is 0.057 IU/ml for anti-D, 0.043 IU/ml for anti-T, 2.693 IU/ml for anti-PT, 2.046 IU/ml for anti-FHA and 2.187 IU/ml for anti-PRN. An agreement between the old and new ELISAs was shown with regards to the two thresholds of clinical relevance for the DI/TE response (0.1 IU/mL and 1.0 IU/mL) and therefore the clinical endpoints and anti-D and anti-T are unchanged. In the absence of a correlate of protection for the pertussis antigens, the anti-PT, anti-FHA and anti-PRN antibody seropositivity endpoints were redefined based on the new assay cut-off.
- 2. Use the SAP template effective since 14-April-2017
- 3. Reflect the protocol amendment 1

The SAP amendment 2 was prepared in order to include the interim analysis of the primary vaccination epoch in the sequence of analysis and in order to reflect the way important protocol deviation will be summarised (Important protocol deviation not leading to elimination will be described using narrative instead of summary table).

# 2. STUDY DESIGN



V = Primary vaccination

BS = Blood Sample

Post-Pri = One month after the third dose of primary vaccination course

Post-Booster = One month after booster vaccination

Protocol waivers or exemptions are not allowed with the exception of immediate safety concerns. Therefore, adherence to the study design requirements, including those specified in the outline of study procedures (Section 5.5 from the protocol), are essential and required for study conduct.

- Experimental design: Phase III, open-label, multi-centric, single-country study with a single group.
- Duration of the study: The intended duration of the study is approximately 16 months, per subject.
  - Epoch 001 (Primary epoch): Primary phase starting at Visit 1 (Day 0) and ending at Visit 4 (Month 4).
  - Epoch 002 (Booster epoch): Booster phase starting at Visit 5 (Month 15) and ending at Visit 6 (Month 16).

Study group: The study group and epochs foreseen in the study are presented in Table 1.

116194 [DTPA-IPV (INFANRIX-IPV)-061] Statistical Analysis Plan Amendment 2 Final

Table 1 Study group and epochs foreseen in the study

| | | | | Epochs |
|---|---|---|---|---|
| Study group | Number of<br>subjects | Age (Min/Max) | Epoch 001<br>(Primary<br>epoch) | Epoch 002 (Booster epoch) |
| DTPa-IPV/Hib<br>Group | ~ 235 | 3 months - 4 months | Х | |
| DTPa-IPV/Hib<br>Group | ~ 235 | 18 months – 19<br>months | | Х |

The study group and treatment foreseen in the study are presented in Table 2.

Table 2 Study group and treatment foreseen in the study

| Treatment name | Vaccine/Product name | Study Group<br>DTPa-IPV/Hib Group |
|------------------|----------------------|-----------------------------------|
| Infanrix-IPV/Hib | DTPa-IPV | X |
| | Hib | X |

- Control: uncontrolled.
- Treatment group and vaccination schedule: All subjects will receive three doses of primary vaccination at 3, 4.5 and 6 months of age and a single dose of booster vaccination at 18 months of age.
  - DTPa-IPV/Hib Group: Subjects who will receive DTPa-IPV/Hib vaccine (Infanrix-IPV/Hib).
- Blinding: This is an open-label study (Refer to Table 3).

Table 3 Blinding of study epochs

| Study Epochs | Blinding |
|---------------------------|----------|
| Epoch 001 (Primary epoch) | open |
| Epoch 002 (Booster epoch) | open |

- Sampling schedule: Two blood samples (approximately 3.5 ml each) will be taken from all subjects: one blood sample will be taken one month after the primary vaccination course (Visit 4) and the second blood sample will be taken one month after the booster vaccination (Visit 6).
- Type of study: This is a self-contained study.
- Data collection: electronic Case Report Form (eCRF).

# 3. OBJECTIVES

# 3.1. Primary objectives

• To assess the immune response to the study vaccine in terms of seroprotection status for diphtheria, tetanus, Hib and poliovirus types 1, 2 and 3 antigens, and in terms of seropositivity to the pertussis antigens, one month after the third dose of primary vaccination.

Refer to Section 4.1 for the definition of the primary endpoint.

# 3.2. Secondary objectives

- To assess the immune response to the study vaccine in terms of seroprotection to diphtheria, tetanus, Hib and poliovirus types 1, 2 and 3 antigens, and in terms of seropositivity to the pertussis antigens, one month after the booster vaccination.
- To assess the immune response to the study vaccine in terms of antibody concentrations or titres against diphtheria, tetanus, Hib, poliovirus types 1, 2 and 3 antigens, and pertussis antigens, one month after the third dose of primary vaccination and one month after the booster vaccination.
- To assess the safety and reactogenicity of the study vaccine in terms of solicited symptoms, unsolicited symptoms and serious adverse events (SAEs).

Refer to Section 4.2 for the definition of the secondary endpoints.

# 4. ENDPOINTS

# 4.1. Primary endpoints

Immunogenicity with respect to components of the study vaccine.

- Anti-diphtheria, anti-tetanus, anti poliovirus types 1, 2 and 3, and anti-PRP seroprotection status, one month after the third dose of primary vaccination.
- Anti- PT, anti-FHA and anti-PRN antibody seropositivity status, one month after the third dose of primary vaccination.

116194 [DTPA-IPV (INFANRIX-IPV)-061] Statistical Analysis Plan Amendment 2 Final

# 4.2. Secondary

- Immunogenicity with respect to components of the study vaccine.
  - Anti-diphtheria, anti-tetanus, anti poliovirus types 1, 2 and 3, and anti-PRP seroprotection status, one month after the booster vaccination.
  - Anti- PT, anti-FHA and anti-PRN antibody seropositivity status, one month after the Booster vaccination
  - Anti-diphtheria, anti-tetanus, anti-poliovirus types 1, 2 and 3, anti-PRP, anti-PT, anti-FHA, anti-PRN antibody concentrations or titres, one month after the third dose of primary vaccination and one month after the booster vaccination.
- Solicited local and general symptoms.
  - Occurrence of solicited local/general symptoms during the 4-day (Days 0-3) follow-up period after each primary vaccination dose and following the booster vaccination.
- Unsolicited adverse events.
  - Occurrence of unsolicited symptoms during the 31-day (Days 0-30) follow-up period after each primary vaccination dose and following the booster vaccination.
- Serious adverse events.
  - Occurrence of SAEs from Dose 1 up to study end.

## 5. ANALYSIS SETS

## 5.1. Definition

## 5.1.1. Total vaccinated cohort (TVC)

The Total vaccinated cohort for the primary epoch will include all subjects who received at least one primary vaccine dose. Thus, the Total vaccinated cohort for analysis of safety of the primary epoch will include all subjects with at least one primary vaccine dose administration documented and the Total vaccinated cohort for analysis of immunogenicity will include vaccinated subjects for whom data concerning primary immunogenicity endpoint measures are available.

The Total vaccinated cohort for the booster epoch will include all subjects who received the booster vaccine dose. Thus, the Total vaccinated cohort for analysis of immunogenicity for the booster epoch will include vaccinated subjects for whom data concerning booster immunogenicity endpoint measures are available.

116194 [DTPA-IPV (INFANRIX-IPV)-061] Statistical Analysis Plan Amendment 2 Final

# 5.1.2. According-to-protocol cohort for analysis of immunogenicity of the primary epoch

The ATP cohort for analysis of immunogenicity of the primary epoch will include all evaluable subjects (i.e. those meeting all eligibility criteria, complying with the procedures and intervals relative to the primary epoch defined in the protocol, with no elimination criteria during the primary epoch of the study) for whom data concerning primary immunogenicity endpoint measures are available. This will include subjects for whom assay results are available for antibodies against at least one study vaccine antigen component one month after Dose 3. The interval between Dose 3 and blood sampling at Visit 4, considered for inclusion of a subject will be 21-48 days.

# 5.1.3. Total vaccinated cohort for the booster epoch

The Total vaccinated cohort for the booster epoch will include all subjects who received the booster dose of study vaccine.

- The TVC for the analysis of safety of booster epoch will include all subjects with booster vaccine dose administration documented.
- The Total vaccinated cohort for analysis of immunogenicity of the booster epoch will include vaccinated subjects for whom data concerning booster immunogenicity endpoint measures are available.

# 5.1.4. According-to-protocol cohort for analysis of immunogenicity of the booster epoch

• The ATP cohort for analysis of immunogenicity of the booster epoch will include all evaluable subjects (i.e. those meeting all eligibility criteria, complying with the procedures and intervals relative to the booster epoch defined in the protocol, with no elimination criteria during the primary and booster epoches of the study) for whom data concerning immunogenicity endpoint measures of booster epoch are available. This will include subjects for whom assay results are available for antibodies against at least one study vaccine antigen component one month after the booster dose of vaccination. The interval between study visits that will be considered for inclusion in the ATP cohort for immunogenicity of booster epoch will be 15–18 months from date of birth to booster vaccination visit and 21-48 days between the booster vaccination visit and the blood sampling at one month post-booster vaccination.

# 5.1.5. Adapted ATP cohort

Adapted ATP cohort for analysis of immunogenicity will be used for tables presenting immunogenicity data from both the primary and booster epoch to indicate that the ATP cohort for analysis of immunogenicity of the primary epoch is used for endpoint at visit 4 (one month post primary) and that the ATP cohort for analysis of immunogenicity of the booster epoch is used for endpoints at visit 6 (one month post booster).

116194 [DTPA-IPV (INFANRIX-IPV)-061] Statistical Analysis Plan Amendment 2 Final

# 5.2. Criteria for eliminating data from Analysis Sets

Elimination codes are used to identify subjects to be eliminated from analysis. Detail is provided below for each sets.

# 5.2.1. Elimination from Total vaccinated cohort (TVC)

Code 1030 (Study vaccine not administered at all) and code 900 (invalid informed consent or fraud data) will be used for identifying subjects eliminated from TVC. The epoch indicator (PR for primary, BO for booster) will be used to indicate the epoch for which data was eliminated.

# 5.2.2. Elimination from ATP cohort for immunogenicity

# 5.2.2.1. Excluded subjects

A subject will be excluded from the ATP cohort for immunogenicity under the following conditions

| Code | Decode => Condition under which the code is used |
|---|---|
| 900 | Questionable subject => Invalid informed consent or fraudulent data. In |
| | case informed consent is obtained retrospectively the subject is not |
| | eliminated. |
| 1030 | Study vaccine dose not administrated at all but subject number allocated => |
| | subjects enrolled but not vaccinated |
| 2010 | Protocol violation (inclusion/exclusion criteria) => ineligible subject: |
| | age outside of (90-120 days) at the time of the first vaccination |
| | Other considerations as stated in section 4.2 – 4.3 in the protocol |
| 2120 | Obvious incoherence or abnormality or error in data => |
| | BS result available while BS not taken |
| | Post booster results below post-primary results for all available assays |
| | tested |

# 5.2.2.2. Right censored Data

| Code | Decode => Condition under which the code is used |
|---|---|
| 1040 | Administration of vaccine(s) forbidden in the protocol => |
| | Use of an investigational or non-registered product (drug or vaccine) other |
| | than the study vaccine used during the study period. |
| | A vaccine not foreseen by the study protocol administered during the period |
| | starting from 30 days before each dose of vaccine and ending 30 days |
| | after*, with the exception of hepatitis B vaccine and other vaccines given as |
| | part of the national immunisation schedule, that are allowed at any time |
| | during the study period. Seasonal or pandemic influenza vaccine can be |
| | given at any time during the study, and according to the Summary of |
| | Product Characteristics and national recommendations. |
| | *In case an emergency mass vaccination for an unforeseen public health |
| | threat (e.g.: a pandemic) is organised by the public health authorities, |
| | outside the routine immunisation program, the time period described above |
| | can be reduced if necessary for that vaccine provided it is licensed and |
| | used according to its SmPC or Prescribing Information and according to the |
| | local governmental recommendations and provided a written approval of |
| 1070 | the Sponsor is obtained. |
| 1070 | Study vaccine dose not administered according to protocol => Route of vaccination is not Intramuscular for DTPa-PV/Hib |
| | Incomplete vaccination course of DTPa-PV/Hib regardless of dropout. |
| | Wrong reconstitution of the DTPa-PV/Hib before injection |
| 1080 | Vaccine temperature deviation => DTPa-PV/Hib vaccine administered |
| 1000 | despite a Good Manufacturing Practices (GMP) no-go temperature |
| | deviation |
| 1090 | Expired vaccine administered=> Subjects who received an expired DTPa- |
| 00.40 | PV/Hib vaccine |
| 2040 | Administration of any medication forbidden by the protocol:=> |
| | Long-acting immune-modifying drugs administered at any time during the |
| | study period (e.g. infliximab). |
| | Use of immunosuppressants or other immune-modifying drugs |
| | administered chronically (i.e., more than 14 days) during the study period. |
| | For corticosteroids, this will mean prednisone ≥0.5 mg/kg/day, or |
| | equivalent. Inhaled and topical steroids are allowed. |
| | Immunoglobulins and/or any blood products administered during the study period |
| 2070 | Concomitant infection not related to the vaccine which may influence |
| | immune response = > Subjects may be eliminated from the ATP cohort for |
| | immunogenicity if, during the study, they incur a condition that has the |
| | capability of altering their immune response (i.e. pertussis infection) or are |
| | confirmed to have an alteration of their initial immune status. |
| 2080 | Non-compliance with vaccination schedule => |
| | Subjects who did not comply with the vaccination interval of 28-62 days |
| | between doses |
| | age outside of (540-570 days) at the time of the booster vaccination |

14-DEC-2017

116194 [DTPA-IPV (INFANRIX-IPV)-061] Statistical Analysis Plan Amendment 2 Final

## 5.2.2.3. Visit-specific censored Data

| Code | Decode => Condition under which the code is used |
|---|---|
| 2090 | Non-compliance with the blood sampling schedule (including wrong and unknown dates) => |
| | Blood sample not collected within 21 days-48 days after the booster dose of the DTPa-PV/Hib vaccine (Visit 6). |
| | Blood sample not collected within 21 days-48 days after the third dose of |
| | the DTPa-PV/Hib vaccine (Visit 4). |
| 2100 | Essential serological data missing => |
| | No serological results at all available post-primary (Visit 4) |
| | No serological results at all available post-booster (Visit 6) or at |

# 5.3. Important protocol deviation not leading to elimination from ATP cohort for immunogenicity

Refer to the protocol deviation management plan for important protocol deviation not leading to elimination from ATP cohort for immunogenicity.

## 6. STATISTICAL ANALYSES

Note that standard data derivation rule and stat methods are described in Section 11 and will not be repeated below.

# 6.1. Demography

# 6.1.1. Analysis of demographics/baseline characteristics planned in the protocol

The analysis of demographics will be performed separately for each epoch:

- The distribution of subjects enrolled among the study centers will be tabulated.
- The number of subjects who withdraw from the study will be tabulated according to the reason for drop-out.
- The deviations from specifications for age and intervals between study visits will be tabulated.

The median, mean, range and standard deviation of age (in weeks) at each vaccine dose will be computed. The median, mean and standard deviation of height in centimeter (cm) and weight in kilograms (kg) at Visit 1 will be computed. The Body Mass Index (BMI) at Visit 1 will also be computed as weight (in kg) / height² (in meters). The gender composition and geographic ancestry will be presented.

14-DEC-2017

116194 [DTPA-IPV (INFANRIX-IPV)-061] Statistical Analysis Plan Amendment 2 Final

## 6.1.2. Additional considerations

The distribution of subjects enrolled among centers and the summary of subjects withdrawal will be generated for the full study on the total vaccinated cohort. All demography summaries will be generated for the TVC and the 2 ATP cohorts. This will include BMI, gender composition and geographic ancestry. Age at first primary vaccination and age at booster vaccination will be computed in weeks.

Number and reason for elimination from each ATP cohort will be tabulated.

# 6.2. Exposure

# 6.2.1. Analysis of exposure planned in the protocol

Not applicable

## 6.2.2. Additional considerations

The number of doses administered will be tabulated.

# 6.3. Immunogenicity

# 6.3.1. Analysis of immunogenicity planned in the protocol

The analysis of immunogenicity will be performed separately for each epoch.

The primary analysis will be based on the ATP cohort for analysis of immunogenicity for both primary and booster epochs. If the percentage of enrolled subjects excluded from this ATP cohort is more than 5%, a second analysis based on the Total vaccinated cohort will be performed on both primary and booster epochs to complement the ATP analysis. All analyses are descriptive.

Where appropriate, at each time-point that a blood-sample result is available:

- Seroprotection rates against diphtheria toxoid, tetanus toxoid, PRP antigen and poliovirus types 1, 2 and 3 antigens (with exact 95% CI) will be calculated.
- Seropositivity rates against PT, FHA and PRN antigens (with exact 95%) will be calculated.
- GMCs/GMTs with 95% CI will be tabulated for antibodies against each antigen.

The distribution of antibody concentrations/titres for each antigen will be displayed using reverse cumulative distribution curves (RCCs).

116194 [DTPA-IPV (INFANRIX-IPV)-061] Statistical Analysis Plan Amendment 2 Final

## Handling of missing data:

• For a given subject and a given immunogenicity measurement, missing or non-evaluable measurements will not be replaced. Therefore, analyses will exclude subjects with missing or non-evaluable measurements.

#### 6.3.2. Additional considerations

The immunogenicity summaries will be generated on the adapted ATP cohort for immunogenicity.

For anti-PRP, the percentage of subjects with antibody concentrations  $\geq 1.0 \,\mu g/ml$  will also be presented with exact 95% CI.

# 6.4. Analysis of safety

# 6.4.1. Analysis of safety planned in the protocol

Analysis of safety relative to the primary epoch will include analysis of safety data collected following administration of the three primary doses of study vaccine. Analysis of safety relative to the booster epoch will include analysis of safety data collected following administration of the booster dose of study vaccine. At this second stage, in order to avoid missing SAEs that have been reported, an SAE summary table including all the events reported during the entire study period will also be generated.

The analysis will be based on the Total vaccinated cohort for both primary and booster epochs. All analyses are descriptive.

- The overall percentage of subjects/doses with at least one local symptom (solicited or unsolicited), with at least one general symptom (solicited or unsolicited) and with any symptom (solicited or unsolicited) during the 4-day (Days 0-3) solicited follow-up period will be tabulated with exact 95% CI after each vaccine dose and overall primary doses. The same calculations will be done for symptoms (solicited or unsolicited) rated as grade 3 in intensity, for symptoms (solicited or unsolicited) leading to medical advice and for symptoms (solicited or unsolicited) assessed as causally related to vaccination.
- The overall percentage of subjects/doses and of subjects reporting each individual solicited local and general symptom during the 4-day (Days 0-3) solicited follow-up period will be tabulated after each vaccine dose and overall primary doses, with exact 95% CI after each vaccine dose and overall primary doses. The same calculations will be done for each individual solicited symptom rated as grade 3 in intensity and for each individual solicited symptom assessed as causally related to vaccination.
- Occurrence of fever will be reported per 0.5°C cumulative increments.

116194 [DTPA-IPV (INFANRIX-IPV)-061] Statistical Analysis Plan Amendment 2 Final

- The verbatim reports of unsolicited AEs will be reviewed by a physician and the signs and symptoms will be coded according to MedDRA. Every verbatim term will be matched with the appropriate Preferred Term. The percentage of subjects with unsolicited AEs occurring within 31-day (Days 0-30) follow-up period after any dose (after primary or booster vaccination) with its exact 95% CI will be tabulated by preferred term. Similar tabulation will be done for unsolicited AEs rated as grade 3, for unsolicited AEs with causal relationship to vaccination and AE(s)/SAE(s) leading to withdrawal from the study.
- The percentage of subjects who receive at least one concomitant medication during the 4-day (Days 0-3) solicited follow-up period and during the entire primary/booster epoch will be tabulated (with exact 95% CI after each vaccine dose and overall.
- Any large injection site reaction (defined as a swelling with a diameter > 50 mm, noticeable diffuse swelling or noticeable increase in limb circumference) after booster vaccination will be described in detail.

SAE(s) will be described in detail.

## Handling of missing data:

- For a given subject and the analysis of solicited symptoms four days postvaccination, missing or non-evaluable measurements will not be replaced. Therefore the analysis of the solicited symptoms based on the TVC will include only vaccinated subjects and doses with documented safety data (i.e., symptom screen completed).
- For analysis of unsolicited AEs, such as SAEs or AEs by primary Medical Dictionary for Regulatory Activities (MedDRA) term, and for the analysis of concomitant medications, all vaccinated subjects will be considered. Subjects, who do not report the event or the concomitant medication, will be considered as subjects without the event or the concomitant medication, respectively.
- For summaries reporting both solicited symptoms and unsolicited AEs, all vaccinated subjects will be considered. Subjects, who do not report the event or the concomitant medication, will be considered as subjects without the event or the concomitant medication, respectively.

## 6.4.2. Additional considerations

The summary of each solicited symptom and unsolicited adverse event will also be done for medically attended symptom/adverse event and for grade 3 causally related.

The percentage of subjects who receive concomitant medication and antipyretic medication during the entire study period will be tabulated for the 31-day (Day 0-30) follow-up period since this is the period planned for collecting concomitant medications.

116194 [DTPA-IPV (INFANRIX-IPV)-061] Statistical Analysis Plan Amendment 2 Final

# 7. ANALYSIS INTERPRETATION

All analyses will be conducted in a descriptive manner.

## 8. CONDUCT OF ANALYSES

Any deviation(s) or change(s) from the original statistical plan outlined in this protocol will be described and justified in the final study report.

# 8.1. Sequence of analyses

The analyses will be performed stepwise:

- A final analysis of the primary epoch will be conducted on all immunogenicity and safety data obtained up to one month after administration of the third primary dose of study vaccine (Visit 4), as soon as the data will be as clean as possible. This will include the analysis of the primary immunogenicity objectives related to the primary epoch and analysis of solicited symptoms and unsolicited adverse events reported within the 4-day (Days 0-3) period and 31-day (Days 0-30) period following the primary vaccination, respectively, and the SAEs reported during the primary epoch.
- Analysis of the booster epoch will be conducted on all cleaned immunogenicity and safety data obtained up to one month after administration of the booster dose of study vaccine (Visit 6). This will include analysis of the secondary immunogenicity objectives related to the booster epoch and analysis of solicited symptoms and unsolicited adverse events reported within the 4-day (Days 0-3) period and 31-day (Days 0-30) period following administration of the booster dose of study vaccine, respectively, and the SAEs reported during the booster epoch. At this second stage, in order to avoid missing SAEs that have been reported, an SAE summary table including all the events reported during the entire study period will also be generated.

# 8.2. Statistical considerations for interim analyses

All analyses will be conducted on final data and therefore no statistical adjustment for interim analyses is required.

| Description | Analysis<br>ID | Disclosure Purpose (IN=internal, CTRS=public posting, SR=study report and public posting) | Dry run<br>review<br>needed<br>(Y/N) | Study Headline<br>Summary<br>(SHS)requiring<br>expedited<br>communication<br>to upper<br>management<br>(Yes/No) | Reference<br>for TFL |
|---|---|---|---|---|---|
| Primary<br>Epoch<br>Analysis | E1_01 | CTRS | Yes | No | TFL TOC |
| Final Analysis | E1_02 | SR and CTRS | Yes | Yes | TFL TOC |

# 8.3. Statistical considerations for interim analyses

The study is descriptive and the interim analysis will be performed on final/clean data. Therefore there is no adjustment for multiplicity resulting from the interim analysis.

## 9. CHANGES FROM PLANNED ANALYSES

Reference to ATP cohort for safety was removed in the description of the ATP cohort for immunogenicity as the ATP cohort for safety was not defined

The Total vaccinated cohort for the booster epoch was defined section 5.1.1

Note that the 2 first secondary endpoints described in the protocol:synopsis refer erroneously to results one month after the Third dose of the primary vaccination as opposed to the secondary endpoints described in the body of the protocol which refer one month post-booster vaccination.

# 10. LIST OF FINAL REPORT TABLES, LISTINGS AND FIGURES

The TFL TOC provides the list of tables/listings and figures needed for the study report. It also identifies the tables eligible for each analyses and their role (synopsis, in-text, post-text, SHS, CTRS,...). Note that all TFL aimed to be included as post-text are noted as post-text even if these are tabulation of individual data such as listing of SAE. The post-text material contain all source material for the study report and accordingly a post-text table may be redundant with an in-text table.

116194 [DTPA-IPV (INFANRIX-IPV)-061] Statistical Analysis Plan Amendment 2 Final

The mock tables referred under column named 'layout' can be found in Section 13 of this SAP.

The following group name will be used in the TFLs, to be in line with the T-domains:

| Group order in tables | Group label in tables | Group definition for footnote |
|---|---|---|
| 1 | DTPa-IPV/Hib | DTPa-IPV/Hib at 3, 4.5, 6 and 18 months of age |

# 11. ANNEX 1 STANDARD DATA DERIVATION RULE AND STATISTICAL METHODS

## 11.1. Statistical Method References

The exact two-sided 95% CIs for a proportion within a group will be the Clopper-Pearson exact CI [Clopper CJ, Pearson ES. The use of confidence or fiducial limits illustrated in the case of binomial. *Biometrika*. 1934;26:404-413].

## 11.2. Standard data derivation

#### 11.2.1. Date derivation

- SAS date derived from a character date: in case day is missing, 15 is used. In case day & month are missing, 30June is used.
- Onset day for an event (ae, medication, vaccination, ...): the onset day is the number of days between the last study vaccination & the onset/start date of the event. This is 0 for an event starting on the same day as a vaccination. See SAS date derived in case the start date of the event is incomplete.

14-DEC-2017

116194 [DTPA-IPV (INFANRIX-IPV)-061] Statistical Analysis Plan Amendment 2 Final

#### 11.2.2. Dose number

- The study dose number is defined in reference to the number of study visits at which vaccination occurred. More specifically dose 1 refers to all vaccines administered at the first vaccination visit while dose 2 corresponds to all vaccinations administered at the second vaccination visit even if this is the first time a product is administered to the subject.
- Relative dose: the relative dose for an event (AE, medication, vaccination) is the most recent study dose given before an event. In case the event takes place on the day a study dose is given, the related dose will be that of the study dose, even if the event actually took place before vaccination. For instance, if an adverse event begins on the day of the study vaccination but prior to administration of the vaccine, it will be assigned to this dose. In case a study dose is not administered and an event occurs after the subsequent study dose (eg 3rd study dose), the relative dose of the event will be study dose associated to the subsequent study dose (eg dose 3).
- The number of doses for a product is the number of time the product was administered to a subject.
- The incidence per dose is the number of vaccination visits at which an event was reported among all vaccination visits.

# 11.2.3. Demography

Age: Age at the reference activity, computed as the number of complete weeks between the date of birth and the reference activity.

Conversion of weight to kg: the following conversion rule is used:

Weight in Kilogram= weight in Pounds / 2.2 + weight in ounces / 35.2

The result is rounded to 2 decimals.

Conversion of height to cm: the following conversion rule is used:

Height in Centimetres = Height in Feet \* 30.48+

Height in Inch \* 2.54

The result is rounded to the unit (ie no decimal).

Conversion of temperature to °C: the following conversion rule is used:

Temperature in °Celsius = ((Temperature in °Fahrenheit -32) \*5)/9

The result is rounded to 1 decimal.

116194 [DTPA-IPV (INFANRIX-IPV)-061] Statistical Analysis Plan Amendment 2 Final

# 11.2.4. Immunogenicity

- A seronegative subject is a subject whose antibody concentration/titre is below the assay cut-off.
- A seropositive subject is a subject whose antibody concentration/titre is greater than or equal to the assay cut-off.
- A seroprotected subject is a subject whose antibody concentration/titre is greater than or equal to the level defining clinical protection. The following seroprotection thresholds are applicable:
  - Anti-diphtheria antibody concentrations  $\geq 0.1 \text{ IU/ml}$ .
  - Anti-tetanus antibody concentrations  $\geq 0.1 \text{ IU/ml}$ .
  - Anti-poliovirus types 1, 2 and 3 antibody titres  $\geq 8$ .
  - Anti-PRP antibody concentrations  $\ge 0.15 \mu g/ml$ .
- The geometric mean titres (GMTs)/geometric mean concentrations (GMCs) calculations will be performed by taking the anti-log of the mean of the log10 titre/concentration transformations. Antibody titres/concentrations below the cut-off of the assay will be given an arbitrary value of half the cut-off for the purpose of GMT/GMC calculation.
- In general, the assay cut-off is the value under which there is no quantifiable result available. For an assay with a specific 'assay cut\_off', numerical immuno result is derived from a character field (rawres):
  - If rawres is 'NEG' or '-' or '(-)', numeric result= assay cut off/2,
  - if rawres is 'POS' or '+' or '(+)', numeric result = assay cut off,
  - if rawres is '< value' and value<=assay cut off, numeric result =assay cut off/2,</li>
  - if rawres is '< value' and value>assay cut off, numeric result =value,
  - if rawres is '> value' and value<assay cut off, numeric result =assay cut off/2,</li>
  - if rawres is '> value' and value>=assay cut off, numeric result =value,
  - if rawres is '<= value' or '>= value' and value<assay cut\_off, numeric result =assay cut\_off/2,</li>
  - if rawres is '<= value' or '>= value' and value>=assay cut\_off, numeric result =value.
  - if rawres is a value < assay cut\_off, numeric result = assay cut\_off/2,</li>
  - if rawres is a value >= assay cut off, numeric result = rawres,
  - else numeric result is left blank.

116194 [DTPA-IPV (INFANRIX-IPV)-061] Statistical Analysis Plan Amendment 2 Final

# 11.2.5. Safety

For analysis of solicited, unsolicited adverse events (such as serious adverse events or adverse events by primary MedDRA term) and for the analysis of concomitant medications, all vaccinated subjects will be considered. Subjects who did not report the event or the concomitant medication will be considered as subjects without the event or the concomitant medication respectively.

The following rules will be used for the analysis of solicited symptoms:

- Subject who didn't document the presence or absence of a solicited symptom
  after one dose will be considered not having that symptom after that dose in the
  analysis done on "administered dose"
- Subjects who documented the absence of a solicited symptom after one dose will be considered not having that symptom after that dose.
- Subjects who documented the presence of a solicited symptom and fully or
  partially recorded daily measurement over the solicited period will be included in
  the summaries at that dose and classified according to their maximum observed
  daily recording over the solicited period.
- Subjects who documented the presence of a solicited symptom after one dose without having recorded any daily measurement will be considered as having that symptom after that dose (at the lowest intensity).
- Intensity of the following solicited AEs will be assessed as described in Table 4 and below

116194 [DTPA-IPV (INFANRIX-IPV)-061] Statistical Analysis Plan Amendment 2 Final

Table 4 Intensity scales to be used by the parent(s)/LAR(s) for solicited symptoms during the solicited follow-up period

| | | Infant |
|---|---|---|
| Adverse Event | Intensity grade | Parameter |
| Pain at injection site | 0 | None |
| - | 1 | Mild: Minor reaction to touch |
| | 2 | Moderate: Cries/protests on touch |
| | 3 | Severe: Cries when limb is moved/spontaneously painful |
| Redness at injection site | | Record greatest surface diameter in mm |
| Swelling at injection site | | Record greatest surface diameter in mm |
| Fever* Record temperature in °C/°F | | |
| Irritability/Fussiness | 0 | Behaviour as usual |
| | 1 | Mild: Crying more than usual/no effect on normal activity |
| | 2 | Moderate: Crying more than usual/interferes with normal activity |
| | 3 | Severe: Crying that cannot be comforted/prevents normal |
| | | activity |
| Drowsiness | 0 | Behaviour as usual |
| | 1 | Mild: Drowsiness easily tolerated |
| | 2 | Moderate: Drowsiness that interferes with normal activity |
| | 3 | Severe: Drowsiness that prevents normal activity |
| Loss of appetite | 0 | Appetite as usual |
| | 1 | Mild: Eating less than usual/no effect on normal activity |
| | 2 | Moderate: Eating less than usual/interferes with normal activity |
| | 3 | Severe: Not eating at all |

<sup>\*</sup>Fever is defined as temperature  $\geq$  37.5°C / 99.5°F for oral, axillary or tympanic route, or  $\geq$  38.0°C / 100.4°F for rectal route.

The maximum intensity of local injection site redness/swelling will be scored at GSK Biologicals as follows:

0 : Absent 1 : ≤ 5 mm

2 :  $> 5 \text{ mm and} \le 20 \text{ mm}$ 

3 : > 20 mm

116194 [DTPA-IPV (INFANRIX-IPV)-061] Statistical Analysis Plan Amendment 2 Final

The maximum intensity of fever will be scored at GSK Biologicals as follows:

# Axillary/Tympanic/Oral

0 :  $< 37.5^{\circ}\text{C} / 99.5^{\circ}\text{F}$ 

1 :  $\geq 37.5^{\circ}\text{C} / 99.5^{\circ}\text{F}$  and

 $\leq 38.0$ °C / 100.4°F

2 : > 38.0°C / 100.4°F and

 $\leq 39.0^{\circ}\text{C} / 102.2^{\circ}\text{F}$ 

3 :  $> 39.0^{\circ}\text{C} / 102.2^{\circ}\text{F}$ 

In case temperature is recorded rectally, a conversion to Axillary temperature will be performed by removing 0.5°C.

Note that for all tables described in this section, the way the percentage of subjects will be derived will depend on the event analysed (see table below for details). As a result, the N value will differ from one table to another.

| Event | N used for deriving % per subject for Vaccination phase | N used for deriving % per dose for<br>Vaccination phase |
|---|---|---|
| Concomitant vaccination | All subjects with study vaccine administered | All study visits with study vaccine administered |
| Solicited<br>general<br>symptom | All subjects with solicited symptoms documented as present or absent for at least one dose. | All doses with solicited symptoms documented as present or absent within 0-3 days post dose |
| Unsolicited symptom | All subjects with study vaccine administered | All study visits with study vaccine administered |
| Concomitant medication | All subjects with study vaccine administered | All study visits with study vaccine administered |

116194 [DTPA-IPV (INFANRIX-IPV)-061] Statistical Analysis Plan Amendment 2 Final

For summaries by MedDRA primary preferred term combining solicited and unsolicited adverse events, solicited adverse events will be coded as per the following MedDRA codes

| Solicited symptom | Lower level term | Corresponding |
|------------------------|------------------|-----------------------|
| | code | Lower level term |
| | | decode |
| Drowsiness | 10013649 | Drowsiness |
| Fever | 10016558 | Fever |
| Irritability/Fussiness | 10022998 | Irritability |
| Loss of appetite | 10003028 | Appetite lost |
| Pain | 10022086 | Injection site pain |
| Redness | | Redness at injection |
| | 10022098 | site |
| Swelling | | Swelling at injection |
| | 10053425 | site |

# 12. ANNEX 2: SUMMARY ON ELIMINATION CODES

Refer to section 5.1.1

# 13. ANNEX 3: STUDY SPECIFIC MOCK TFL

The following draft study specific mock TFLs will be used.

The data display, title and footnote are for illustration purpose and will be adapted to the study specificity as indicated in the TFL TOC.

These templates were copied from recent studies. Note that there may be few changes between the study specific SAP mock TFL and the final TFLs. These editorial/minor changes will not lead to a SAP amendment.

116194 [DTPA-IPV (INFANRIX-IPV)-061] Statistical Analysis Plan Amendment 2 Final

Template 1 Number of subjects enrolled by center - TVC

| | Combo group | Control group | | Total |
|--------|-------------|---------------|-----|-------|
| Center | n | n | n | % |
| PPD | 20 | 21 | 41 | 9.1 |
| PPD | 27 | 28 | 55 | 12.2 |
| PPD | 7 | 7 | 14 | 3.1 |
| PPD | 16 | 16 | 32 | 7.1 |
| PPD | 27 | 26 | 53 | 11.8 |
| PPD | 26 | 26 | 52 | 11.5 |
| PPD | 25 | 25 | 50 | 11.1 |
| PPD | 23 | 24 | 47 | 10.4 |
| PPD | 22 | 22 | 44 | 9.8 |
| PPD | 24 | 25 | 49 | 10.9 |
| PPD | 7 | 7 | 14 | 3.1 |
| All | 224 | 227 | 451 | 100 |

<group description >

n = number of subjects included in each group or in total for a given center or for all centers

All = sum of all subjects in each group or in total (sum of all groups)

 $% = n/AII \times 100$ 

Template 2 Number of subjects vaccinated, completed and withdrawn with reason for withdrawal at Visit 3 - TVC

| | HRV Liq | HRV | Total |
|---|---|---|---|
| | | LYO | |
| Number of subjects vaccinated | 300 | 300 | 1200 |
| Number of subjects completed | 298 | 297 | 1193 |
| Number of subjects withdrawn | 2 | 3 | 7 |
| Reasons for withdrawal : | | | |
| Serious Adverse Event | 0 | 1 | 1 |
| Non-serious adverse event | 0 | 0 | 0 |
| Protocol violation | 0 | 0 | 0 |
| Consent withdrawal (not due to an adverse event) | 1 | 2 | 4 |
| Migrated/moved from study area | 1 | 0 | 2 |
| Lost to follow-up (subjects with incomplete vaccination course) | 0 | 0 | 0 |
| Lost to follow-up (subjects with complete vaccination course) | 0 | 0 | 0 |
| Others | 0 | 0 | 0 |

HRV LIQ = HRV vaccine liquid formulation

HRV LYO = HRV vaccine HRV Lyophilised formulation

Vaccinated = number of subjects who were vaccinated in the study

Completed = number of subjects who completed study visit 3

Withdrawn = number of subjects who did not come for study visit 3

116194 [DTPA-IPV (INFANRIX-IPV)-061] Statistical Analysis Plan Amendment 2 Final

Template 3 Number of subjects at each visit and list of withdrawn subjects (TVC)

| Group | VISIT | N | Withdrawn<br>Subject numbers | Reason for withdrawal |
|---|---|---|---|---|
| HRV Liq | VISIT 1 | 508 | • | |
| | - | | no. PP | CONSENT WITHDRAWAL |
| | | | Ino PP | CONSENT WITHDRAWAL |
| | | | no PPD | CONSENT WITHDRAWAL |
| | | | no. PPD | CONSENT WITHDRAWAL |
| | VISIT 2 | 504 | | |
| | - | | no. PPD | CONSENT WITHDRAWAL |
| | | | no. PPD | CONSENT WITHDRAWAL |
| | | | no. PPD | SERIOUS ADVERSE EXPERIENCE |
| | VISIT 3 | 501 | | |
| | | | no. P | MIGRATION FROM STUDY AREA |
| | | | no. PP | CONSENT WITHDRAWAL |
| | | | no. PP | MIGRATION FROM STUDY AREA |
| | | | no. PP | CONSENT WITHDRAWAL |
| | | | no. PP | MIGRATION FROM STUDY AREA |
| | | | no. PP | MIGRATION FROM STUDY AREA |
| | | | no. PPD | CONSENT WITHDRAWAL |
| | | | no. PPD | MIGRATION FROM STUDY AREA |
| | | | no. PPD | MIGRATION FROM STUDY AREA |
| | VISIT 4 | 492 | | |
| HRV Lyo | VISIT 1 | 257 | | |
| | | | no. PP | PROTOCOL VIOLATION |
| | | | no. PPD | CONSENT WITHDRAWAL |
| | VISIT 2 | 255 | | |
| | | | no. PPD | CONSENT WITHDRAWAL |
| | VISIT 3 | 254 | | |
| | | | no. PP | MIGRATION FROM STUDY AREA |
| | | | no. PP | LOST TO FOLLOW-UP |
| | | | no. PP | LOST TO FOLLOW-UP |
| | | | no. PP | CONSENT WITHDRAWAL |
| | | | no. PP | MIGRATION FROM STUDY AREA |
| | | | no. PPD | LOST TO FOLLOW-UP |
| | | | no. PPD | ADVERSE EXPERIENCE |
| | VISIT 4 | 247 | | |

116194 [DTPA-IPV (INFANRIX-IPV)-061] Statistical Analysis Plan Amendment 2 Final

Template 4 Number of subjects enrolled into the study as well as the number of subjects excluded from ATP analyses with reasons for exclusion

| | | To | tal | | H | IRV LI | Q | HRV LYO | | |
|---|---|---|---|---|---|---|---|---|---|---|
| Title | N | n | S | % | N | n | S | N | n | s |
| Total enrolled cohort | 1200 | | | | 300 | | | 300 | | |
| TVC | 1200 | | | 100 | 300 | | | 300 | | |
| Administration of vaccine(s) forbidden in | | 2 | 2 | | | 0 | 0 | | 0 | 0 |
| the protocol | | | | | | | | | | |
| (code 1040) | | | | | | | | | | |
| Study vaccine dose not administered | | 73 | 73 | | | 23 | 23 | | 16 | 16 |
| according to protocol (code 1070) | | | | | | | | | | |
| Initially seropositive or unknown anti- | | 10 | 11 | | | 3 | 3 | | 1 | 1 |
| rotavirus IgA antibody on day of dose 1 | | | | | | | | | | |
| (code 1500) | | | | | | | | | | |
| Protocol violation (inclusion/exclusion | | 1 | 1 | | | 1 | 1 | | 0 | 0 |
| criteria) | | | | | | | | | | |
| (code 2010) | | | | | | | | | | |
| Administration of any medication forbidden | | 1 | 1 | | | 0 | 0 | | 1 | 1 |
| by the protocol (code 2040) | | | | | | | | | | |
| Underlying medical condition forbidden by | | 1 | 1 | | | 0 | 0 | | 0 | 0 |
| the protocol | | | | | | | | | | |
| (code 2050) | | | | | | | | | | |
| Concomitant infection not related to the | | 0 | 1 | | | 0 | 0 | | 0 | 1 |
| vaccine which may influence immune | | | | | | | | | | |
| response (code 2070) | | | | | | | | | | |
| Non compliance with vaccination schedule | | 14 | 16 | | | 6 | 7 | | 3 | 4 |
| (including wrong and unknown dates) | | | | | | | | | | |
| (code 2080) | | | | | | | | | | |
| Non compliance with blood sampling | | 12 | 16 | | | 3 | 5 | | 4 | 5 |
| schedule (including wrong and unknown | | | | | | | | | | |
| dates) | | | | | | | | | | |
| (code 2090) | | | | | | | | | | |
| Essential serological data missing (code | | 87 | 95 | | | 20 | 22 | | 23 | 26 |
| 2100) | | | | | | | | | | |
| Subjects with incomplete study vaccination | | 1 | 1 | | | 0 | 0 | | 0 | 0 |
| schedule but with post serological result | | | | | | | | | | |
| (code 2500) | | | | | | | | | | |
| ATP | 998 | | <u></u> | 83.2 | 244 | | | 252 | | |

HRV LIQ = HRV vaccine liquid formulation Lot C HRV LYO = HRV vaccine HRV Lyophilised formulation

Note: Subjects may have more than one elimination code assigned

n = number of subjects with the elimination code assigned excluding subjects who have been assigned a lower elimination code number

s = number of subjects with the elimination code assigned

<sup>% =</sup> percentage of subjects in the per protocol set (ATP) relative to the TVC (ES)

116194 [DTPA-IPV (INFANRIX-IPV)-061] Statistical Analysis Plan Amendment 2 Final

Template 5 Deviations from specifications for age and intervals between study visits - TVC

| | | Age | PRE-Dose:1 | Dose:1 | -Dose:2 | Dose:2 | -PII(M2) |
|---|---|---|---|---|---|---|---|
| Group | | Protocol | Protocol | Protocol | Adapted | Protocol | Adapted |
| • | | from 10 to 17 | from 0 to 0 days | from 30 to 48 | from 21 to 48 | from 30 to 48 | |
| | | weeks | - | days | days | days | days |
| HRV<br>LIQ | N | 300 | 300 | 300 | 300 | 291 | 291 |
| | n | 1 | 1 | 8 | 7 | 4 | 4 |
| | % | 0.3 | 0.3 | 2.7 | 2.3 | 1.4 | 1.4 |
| | range | 9 to 17 | 0 to 9 | 27 to 76 | 27 to 76 | 30 to 56 | 30 to 56 |
| HRV<br>LYO | N | 300 | 300 | 299 | 299 | 289 | 289 |
| | n | 0 | 2 | 4 | 4 | 5 | 3 |
| | % | 0.0 | 0.7 | 1.3 | 1.3 | 1.7 | 1.0 |
| | range | 10 to 16 | 0 to 3 | 30 to 61 | 30 to 61 | 28 to 61 | 28 to 61 |

HRV LIQ = HRV vaccine liquid formulation Lot A

HRV LIQ = HRV vaccine liquid formulation Lot B

HRV LIQ = HRV vaccine liquid formulation Lot C

HRV LYO = HRV vaccine HRV Lyophilised formulation

PRE = pre-vaccination

PII (M2) = blood sample taken one month after Dose 2 of the HRV vaccine (Visit 3)

Adapted = interval used for defining the ATP cohorts for immunogenicity

N = total number of subjects with available results

n/% = number / percentage of subjects with results outside of the interval

range = minimum-maximum for age and intervals

116194 [DTPA-IPV (INFANRIX-IPV)-061] Statistical Analysis Plan Amendment 2 Final

Template 6 Summary of demographic characteristics (ATP cohort for Immunogenicity)

| | | HRV LIC | | HRV L | - | Total | |
|---|---|---|---|---|---|---|---|
| | | N = 244 | | N = 252 | | N = 998 | |
| Characteristics | Parameters or | Value | % | Value | % | Value | % |
| | Categories | or n | | or n | | or n | |
| Age at Dose 1 | Mean | 11.5 | - | 11.6 | - | 11.6 | - |
| of HRV vaccine | SD | 1.19 | - | 1.20 | - | 1.22 | - |
| (weeks) | Median | 11.0 | - | 11.0 | - | 11.0 | - |
| | Minimum | 10 | - | 10 | - | 10 | - |
| | Maximum | 15 | - | 16 | - | 17 | - |
| Age at Dose 2 | Mean | 16.5 | - | 16.7 | - | 16.6 | - |
| of HRV vaccine | SD | 1.37 | - | 1.34 | - | 1.40 | - |
| (weeks) | Median | 16.0 | - | 17.0 | - | 17.0 | - |
| | Minimum | 14 | - | 14 | - | 14 | - |
| | Maximum | 20 | - | 21 | - | 22 | - |
| Gender | Female | 120 | 49.2 | 120 | 47.6 | 483 | 48.4 |
| | Male | 124 | 50.8 | 132 | 52.4 | 515 | 51.6 |
| Ethnicity | American Hispanic or Latino | 1 | 0.4 | 0 | 0.0 | 3 | 0.3 |
| - | Not American Hispanic or Latino | 243 | 99.6 | 252 | 100.0 | 995 | 99.7 |
| Race | African heritage / African American | 1 | 0.4 | 0 | 0.0 | 2 | 0.2 |
| | American Indian or Alaskan native | 0 | 0.0 | 0 | 0.0 | 0 | 0.0 |
| | Asian - central/south Asian heritage | 0 | 0.0 | 0 | 0.0 | 0 | 0.0 |
| | Asian - east Asian heritage | 0 | 0.0 | 0 | 0.0 | 0 | 0.0 |
| | Asian - Japanese heritage | 0 | 0.0 | 0 | 0.0 | 0 | 0.0 |
| | Asian - south east Asian heritage | 0 | 0.0 | 0 | 0.0 | 0 | 0.0 |
| | Native Hawaiian or other pacific islander | 0 | 0.0 | 0 | 0.0 | 0 | 0.0 |
| | White - Arabic / north African heritage | 2 | 8.0 | 0 | 0.0 | 2 | 0.2 |
| | White - Caucasian / European heritage | 240 | 98.4 | 247 | 98.0 | 984 | 98.6 |
| | Other | 1 | 0.4 | 5 | 2.0 | 10 | 1.0 |
| Height at Visit | Mean | 60.7 | - | 60.6 | - | 60.5 | - |
| 1 (cm) | SD | 2.32 | - | 2.22 | - | 2.32 | _ |
| , | Median | 61.0 | - | 61.0 | - | 61.0 | _ |
| | Unknown | 2 | - | 0 | - | 3 | _ |
| Weight at Visit | Mean | 6.2 | - | 6.1 | - | 6.1 | - |
| 1 (kg) | SD | 0.77 | - | 0.75 | - | 0.76 | - |
| · •/ | Median | 6.2 | - | 6.1 | - | 6.1 | - |
| BMI at Visit 1 | Mean | 16.7 | - | 16.7 | - | 16.6 | - |
| (kg/m²) | SD | 1.46 | - | 1.46 | - | 1.47 | - |
| \ J/ | Median | 16.5 | - | 16.7 | - | 16.5 | - |
| | Unknown | 2 | - | 0 | _ | 3 | _ |

HRV LIQ = HRV vaccine liquid formulation Lot A

HRV LIQ = HRV vaccine liquid formulation Lot B

HRV LIQ = HRV vaccine liquid formulation Lot C

HRV LYO = HRV vaccine HRV Lyophilised formulation

N = total number of subjects

n (%) = number / percentage of subjects in a given category

Value = value of the considered parameter

SD = standard deviation

116194 [DTPA-IPV (INFANRIX-IPV)-061] Statistical Analysis Plan Amendment 2 Final

## **Template 7** Study population (TVC)

| Study population (Total vaccinated cohort) | | |
|---|---|---|
| Number of subjects | Combo group | Control group |
| Planned, N | 225 | 225 |
| Randomised, N (Total Vaccinated Cohort) | 224 | 227 |
| Completed, n (%) | 224 (100) | 227 (100) |
| Demographics | Combo group | Control group |
| N (Total Vaccinated Cohort) | 224 | 227 |
| Females :Males | 97:127 | 115:112 |
| Mean Age, weeks (SD) | 8.8 (1.1) | 8.8 (1.1) |
| Median Age, weeks (minimum, maximum) | 9 (7, 11) | 9 (7, 11) |
| Most frequent race: Asian - East Asian Heritage, n (%) | 224 (100) | 226 (99.6) |

Combo group = Subjects received DTPa-IPV/Hib vaccine as a single injection at 2, 4 and 6 months of age

Control group = Subjects received DTPa-IPV and Hib vaccines at different injection sites at 2, 4 and 6 months of age

N = Total number of subjects enrolled in the study

n/% = Number/percentage of subjects in a given category

SD = Standard Deviation

MeaAge = Age calculated from Date of birth to first study vaccination

Template 8 Anti-rotavirus IgA antibody GMC and seropositivity rates – ATP cohort for Immunogenicity

| | Timing | ≥<br> N n | ≥ 20 U | ≥ 20 U/ml | | | GMC (U/r | GMC (U/ml) | |
|---|---|---|---|---|---|---|---|---|---|
| Group | | | | | 95% CI | | | 95% CI | |
| | | | n | % | LL | UL | value | LL | UL |
| HRV LIQ | PRE | 244 | 0 | 0.0 | 0.0 | 1.5 | <20 | - | - |
| | PII(M2) | 244 | 206 | 84.4 | 79.3 | 88.7 | 324.4 | 253.4 | 415.3 |
| HRV LYO | PRE | 252 | 0 | 0.0 | 0.0 | 1.5 | <20 | - | - |
| | PII(M2) | 252 | 228 | 90.5 | 86.2 | 93.8 | 331.8 | 265.0 | 415.4 |

HRV LIQ = HRV vaccine liquid formulation Lot C LIQPOOL = Pooled HRV vaccine liquid formulation

HRV LYO = HRV vaccine HRV Lyophilised formulation

N = number of subjects with available results

n (%) = number/percentage of subjects with concentration above the cut-off

95% CI = 95% Confidence Interval; L.L =Lower limit; U.L = upper limit

Pre = pre-vaccination

PII (M2) = blood sample taken one month after Dose 2 of HRV vaccine (Visit 3)

116194 [DTPA-IPV (INFANRIX-IPV)-061] Statistical Analysis Plan Amendment 2 Final

Template 9 Reverse cumulative distribution curve for anti-rotavirus IgA antibody concentrations at Visit 3 - ATP cohort for Immunogenicity


116194 [DTPA-IPV (INFANRIX-IPV)-061] Statistical Analysis Plan Amendment 2 Final

Template 10 Number and percentage of subjects who received study vaccine doses - TVC

| | | | ' LIQ<br>300 | HRV<br>N = | | | tal<br>1200 |
|---|---|---|---|---|---|---|---|
| VACCINE | Total number of doses received | n | % | n | % | n | % |
| Pediarix | 1 | 0 | 0.0 | 1 | 0.3 | 3 | 0.3 |
| | 2 | 300 | 100 | 299 | 99.7 | 1197 | 99.8 |
| | 3 | | | | | | |
| Any | Any | 300 | 100 | 300 | 100 | 1200 | 100 |
| Hiberix | 1 | 0 | 0.0 | 1 | 0.3 | 3 | 0.3 |
| | 2 | 300 | 100 | 299 | 99.7 | 1197 | 99.8 |
| | 3 | | | | | | |
| Any | Any | 300 | 100 | 300 | 100 | 1200 | 100 |
| Prevnar | 1 | 0 | 0.0 | 1 | 0.3 | 3 | 0.3 |
| | 2 | 300 | 100 | 299 | 99.7 | 1197 | 99.8 |
| | 3 | | | | | | |
| Any ON COAD | Any | 300 | 100 | 300 | 100 | 1200 | 100 |

HRV LIQ = HRV vaccine Liquid formulation lot A HRV LIQ = HRV vaccine Liquid formulation lot B

HRV LIQ = HRV vaccine Liquid formulation lot C HRV LYO = HRV vaccine HRV Lyophilised formulation

N = number of subjects in each group or in total included in the considered cohort

n (%) = number/percentage of subjects receiving the specified total number of doses

Any = number and percentage of subjects receiving at least one dose

Template 11 Compliance in returning symptom sheets - TVC

| Dose | GROUP | Number | Doses | Number | Compliance |
|---|---|---|---|---|---|
| | | of doses | NOT according to protocol | of general SS | % general SS |
| 1 | HRV LIQ | 298 | 10 | 298 | 100 |
| | HRV LIQ | 302 | 7 | 302 | 100 |
| | HRV LIQ | 300 | 6 | 300 | 100 |
| | LIQPOOL | 900 | 23 | 900 | 100 |
| | HRV LYO | 300 | 6 | 299 | 99.7 |
| 2 | HRV LIQ | 297 | 12 | 296 | 99.7 |
| | HRV LIQ | 301 | 6 | 301 | 100 |
| | HRV LIQ | 300 | 13 | 299 | 99.7 |
| | LIQPOOL | 898 | 31 | 896 | 99.8 |
| | HRV LYO | 299 | 9 | 297 | 99.3 |
| Total | HRV LIQ | 595 | 22 | 594 | 99.8 |
| | HRV LIQ | 603 | 13 | 603 | 100 |
| | HRV LIQ | 600 | 19 | 599 | 99.8 |
| | LIQPOOL | 1798 | 54 | 1796 | 99.9 |
| | HRV LYO | 599 | 15 | 596 | 99.5 |

HRV LIQ = HRV vaccine liquid formulation Lot A

HRV LIQ = HRV vaccine liquid formulation Lot B

HRV LIQ = HRV vaccine liquid formulation Lot C

LIQPOOL = Pooled HRV vaccine liquid formulation

HRV LYO = HRV vaccine HRV Lyophilised formulation

SS = Symptom sheets used for the collection of solicited AEs

Compliance % = (number of doses with symptom sheet return / number of administered doses) X 100

Doses not according to protocol = number of doses with regurgitation or vomiting

116194 [DTPA-IPV (INFANRIX-IPV)-061] Statistical Analysis Plan Amendment 2 Final

Template 12 Incidence and nature of grade 3 symptoms (solicited and unsolicited) reported during the 4-day (Days 0-3) period after vaccination following each dose and overall (Total vaccinated cohort)

| | | | Ar | ny syn | nptom | | Ge | ener | al sy | mpto | oms | | Loc | al syn | nptom | IS |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | | | 959 | % CI | | | | 95 | % CI | | | _ | 959 | % CI |
| | Group | N | n | % | LL | UL | N | n | % | LL | UL | N | n | % | LL | UL |
| Dose 2 | Combo group | 224 | 18 | 8.0 | 4.8 | 12.4 | 224 | 7 | 3.1 | 1.3 | 6.3 | 224 | 12 | 5.4 | 2.8 | 9.2 |
| | Control group | 227 | 15 | 6.6 | 3.7 | 10.7 | 227 | 6 | 2.6 | 1.0 | 5.7 | 227 | 11 | 4.8 | 2.4 | 8.5 |
| Dose 4 | Combo group | 224 | 29 | 12.9 | 8.8 | 18.1 | 224 | 6 | 2.7 | 1.0 | 5.7 | 224 | 26 | 11.6 | 7.7 | 16.5 |
| | Control group | 227 | 29 | 12.8 | 8.7 | 17.8 | 227 | 9 | 4.0 | 1.8 | 7.4 | 227 | 22 | 9.7 | 6.2 | 14.3 |
| Dose 6 | Combo group | 224 | 25 | 11.2 | 7.4 | 16.0 | 224 | 8 | 3.6 | 1.6 | 6.9 | 224 | 18 | 8.0 | 4.8 | 12.4 |
| | Control group | 227 | 19 | 8.4 | 5.1 | 12.8 | 227 | 2 | 0.9 | 0.1 | 3.1 | 227 | 18 | 7.9 | 4.8 | 12.2 |
| Overall/dose | Combo group | 672 | 72 | 10.7 | 8.5 | 13.3 | 672 | 21 | 3.1 | 1.9 | 4.7 | 672 | 56 | 8.3 | 6.4 | 10.7 |
| | Control group | 681 | 63 | 9.3 | 7.2 | 11.7 | 681 | 17 | 2.5 | 1.5 | 4.0 | 681 | 51 | 7.5 | 5.6 | 9.7 |
| Overall/subject | Combo group | 224 | 60 | 26.8 | 21.1 | 33.1 | 224 | 21 | 9.4 | 5.9 | 14.0 | 224 | 44 | 19.6 | 14.7 | 25.5 |
| ,<br> | Control group | 227 | 47 | 20.7 | 15.6 | 26.6 | 227 | 14 | 6.2 | 3.4 | 10.1 | 227 | 39 | 17.2 | 12.5 | 22.7 |

Combo group = Subjects received DTPa-IPV/Hib vaccine as a single injection at 2, 4 and 6 months of age

Control group = Subjects received DTPa-IPV and Hib vaccines at different injection sites at 2, 4 and 6 months of age For each dose and overall/subject:

N = number of subjects with at least one administered dose

n/% = number/percentage of subjects presenting at least one type of symptom whatever the study vaccine administered

For overall/dose:

N = number of administered doses

n/% = number/percentage of doses followed by at least one type of symptom whatever the study vaccine administered 95% CI = exact 95% confidence interval, LL = Lower Limit, UL = Upper Limit

Dose 2, 4 and 6 are the doses where subjects has received study vaccine - DTPa-IPV/Hib vaccine in Combo group and DTPa-IPV and Hib in Control group

116194 [DTPA-IPV (INFANRIX-IPV)-061] Statistical Analysis Plan Amendment 2 Final

Template 13 Incidence of solicited local symptoms reported during the 4-day (Days 0-3) period after vaccination following each dose and overall (Total vaccinated cohort)

| | | | ( | Combo | group | | | ( | Control | group | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | | | | % CI | | | | | i % CI |
| Symptom | Туре | N | n | % | LL | UL | N | n | % | LL | UL |
| | | | | Dos | e 2 | | | | | | |
| Pain | All | 224 | 108 | 48.2 | 41.5 | 55.0 | 227 | 113 | 49.8 | 43.1 | 56.5 |
| | Grade 3 | 224 | 5 | 2.2 | 0.7 | 5.1 | 227 | 8 | 3.5 | 1.5 | 6.8 |
| Redness (mm) | All | 224 | 133 | 59.4 | 52.6 | 65.9 | 227 | 119 | 52.4 | 45.7 | 59.1 |
| | >20 | 224 | 4 | 1.8 | 0.5 | 4.5 | 227 | 3 | 1.3 | 0.3 | 3.8 |
| Swelling (mm) | All | 224 | 65 | 29.0 | 23.2 | 35.4 | 227 | 64 | 28.2 | 22.4 | 34.5 |
| | >20 | 224 | 5 | 2.2 | 0.7 | 5.1 | 227 | 2 | 0.9 | 0.1 | 3.1 |
| | · | | | Dos | | | | | | | |
| Pain | All | 224 | 81 | 36.2 | 29.9 | 42.8 | 227 | 88 | 38.8 | 32.4 | 45.4 |
| | Grade 3 | 224 | 3 | 1.3 | 0.3 | 3.9 | 227 | 3 | 1.3 | 0.3 | 3.8 |
| Redness (mm) | All | 224 | 131 | 58.5 | 51.7 | 65.0 | 227 | 124 | 54.6 | 47.9 | 61.2 |
| | >20 | 224 | 20 | 8.9 | 5.5 | 13.5 | 227 | 18 | 7.9 | 4.8 | 12.2 |
| Swelling (mm) | All | 224 | 85 | 37.9 | 31.6 | 44.7 | 227 | 78 | 34.4 | 28.2 | 40.9 |
| | >20 | 224 | 9 | 4.0 | 1.9 | 7.5 | 227 | 4 | 1.8 | 0.5 | 4.5 |
| | | | | Dos | e 6 | | | | | | |
| Pain | All | 224 | 87 | 38.8 | 32.4 | 45.6 | 227 | 78 | 34.4 | 28.2 | 40.9 |
| | Grade 3 | 224 | 1 | 0.4 | 0.0 | 2.5 | 227 | 3 | 1.3 | 0.3 | 3.8 |
| Redness (mm) | All | 224 | 128 | 57.1 | 50.4 | 63.7 | 227 | 122 | 53.7 | 47.0 | 60.4 |
| | >20 | 224 | 14 | 6.3 | 3.5 | 10.3 | 227 | 14 | 6.2 | 3.4 | 10.1 |
| Swelling (mm) | All | 224 | 96 | 42.9 | 36.3 | 49.6 | 227 | 88 | 38.8 | 32.4 | 45.4 |
| | >20 | 224 | 6 | 2.7 | 1.0 | 5.7 | 227 | 7 | 3.1 | 1.2 | 6.3 |
| | | | | Overall | l/dose | | | | | | |
| Pain | All | 672 | 276 | 41.1 | 37.3 | 44.9 | 681 | 279 | 41.0 | 37.2 | 44.8 |
| | Grade 3 | 672 | 9 | 1.3 | 0.6 | 2.5 | 681 | 14 | 2.1 | 1.1 | 3.4 |
| Redness (mm) | All | 672 | 392 | 58.3 | 5 | 62.1 | 681 | 365 | 53.6 | 49.8 | 57.4 |
| | >20 | 672 | 38 | 5.7 | 4.0 | 7.7 | 681 | 35 | 5.1 | 3.6 | 7.1 |
| Swelling (mm) | All | 672 | 246 | 36.6 | 33.0 | 40.4 | 681 | 230 | 33.8 | 30.2 | 37.5 |
| | >20 | 672 | 20 | 3.0 | 1.8 | 4.6 | 681 | 13 | 1.9 | 1.0 | 3.2 |
| | | | ( | Overall/s | subject | | | | | | |
| Pain | All | 224 | 143 | 63.8 | 57.2 | 70.1 | 227 | 146 | 64.3 | 57.7 | 70.5 |
| | Grade 3 | 224 | 9 | 4.0 | 1.9 | 7.5 | 227 | 12 | 5.3 | 2.8 | 9.1 |
| Redness (mm) | All | 224 | 177 | 79.0 | 73.1 | 84.2 | 227 | 167 | 73.6 | 67.3 | 79.2 |
| | >20 | 224 | 29 | 12.9 | 8.8 | 18.1 | 227 | 26 | 11.5 | 7.6 | 16.3 |
| Swelling (mm) | All | 224 | 130 | 58.0 | 51.3 | 64.6 | 227 | 121 | 53.3 | 46.6 | 59.9 |
| | >20 | 224 | 15 | 6.7 | 3.8 | 10.8 | 227 | 11 | 4.8 | 2.4 | 8.5 |

Combo group = Subjects received DTPa-IPV/Hib vaccine as a single injection at 2, 4 and 6 months of age

Control group = Subjects received DTPa-IPV and Hib vaccines at different injection sites at 2, 4 and 6 months of age For each dose and overall/subject:

N = number of subjects with at least one documented dose

n/% = number/percentage of subjects reporting the symptom at least once

For Overall/dose:

N = number of documented doses

n/% = number/percentage of doses followed by at least one type of symptom

95%CI = Exact 95% confidence interval; LL = lower limit, UL = upper limit

Dose 2, 4 and 6 are the doses where subjects has received study vaccine - DTPa-IPV/Hib vaccine in Combo group and DTPa-IPV and Hib in Control group

Grade 3 pain refers to severe significant pain at rest. Prevents normal every day activities.

116194 [DTPA-IPV (INFANRIX-IPV)-061] Statistical Analysis Plan Amendment 2 Final

Template 14 Percentage of doses with solicited general symptom including those rated grade 3 in intensity and those assessed as related to vaccination during the 8-day (Day 1 to Day 8) follow-up period, for each dose in the pooled HRV vaccine liquid formulation group and the HRV vaccine HRV Lyophilised formulation group - TVC

| | | LIQPO | OOL | | | | HRV I | LYO | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | | | 95 % | CI | | | | 95 % | CI |
| Symptom | Туре | N | n | % | LL | UL | N | n | % | LL | UL |
| Dose 1 | | | | | | | | | | | |
| Cough/runny nose | All | 900 | 233 | 25.9 | 23.1 | 28.9 | 300 | 79 | 26.3 | 21.4 | 31.7 |
| | Grade 3 | 900 | 2 | 0.2 | 0.0 | 0.8 | 300 | 4 | 1.3 | 0.4 | 3.4 |
| | Related | 900 | 187 | 20.8 | 18.2 | 23.6 | 300 | 64 | 21.3 | 16.8 | 26.4 |
| Diarrhoea | All | 900 | 25 | 2.8 | 1.8 | 4.1 | 300 | 4 | 1.3 | 0.4 | 3.4 |
| | Grade 3 | 900 | 7 | 0.8 | 0.3 | 1.6 | 300 | 1 | 0.3 | 0.0 | 1.8 |
| | Related | 900 | 25 | 2.8 | 1.8 | 4.1 | 300 | 3 | 1.0 | 0.2 | 2.9 |
| Fever(°C) | All | 900 | 179 | 19.9 | 17.3 | 22.6 | 300 | 68 | 22.7 | 18.1 | 27.8 |
| , , | Grade 3 | 900 | 2 | 0.2 | 0.0 | 0.8 | 300 | 0 | 0.0 | 0.0 | 1.2 |
| | Related | 900 | 174 | 19.3 | 16.8 | 22.1 | 300 | 67 | 22.3 | 17.7 | 27.5 |
| Irritability | All | 900 | 629 | 69.9 | 66.8 | 72.9 | 300 | 207 | 69.0 | 63.4 | 74.2 |
| • | Grade 3 | 900 | 38 | 4.2 | 3.0 | 5.7 | 300 | 12 | 4.0 | 2.1 | 6.9 |
| | Related | 900 | 607 | 67.4 | 64.3 | 70.5 | 300 | 201 | 67.0 | 61.4 | 72.3 |
| Loss of appetite | All | 900 | 231 | 25.7 | 22.8 | 28.7 | 300 | 67 | 22.3 | 17.7 | 27.5 |
| • • | Grade 3 | 900 | 1 | 0.1 | 0.0 | 0.6 | 300 | 1 | 0.3 | 0.0 | 1.8 |
| | Related | 900 | 220 | 24.4 | 21.7 | 27.4 | 300 | 63 | 21.0 | 16.5 | 26.1 |
| Vomiting | All | 900 | 136 | 15.1 | 12.8 | 17.6 | 300 | 55 | 18.3 | 14.1 | 23.2 |
| · · | Grade 3 | 900 | 25 | 2.8 | 1.8 | 4.1 | 300 | 11 | 3.7 | 1.8 | 6.5 |
| | Related | 900 | 127 | 14.1 | 11.9 | 16.6 | 300 | 51 | 17.0 | 12.9 | 21.7 |
| Dose 2 | | | | 1 | | | | | | | |
| Cough/runny nose | All | 898 | 291 | 32.4 | 29.4 | 35.6 | 299 | 109 | 36.5 | 31.0 | 42.2 |
| 0 , | Grade 3 | 898 | 8 | 0.9 | 0.4 | 1.7 | 299 | 2 | 0.7 | 0.1 | 2.4 |
| | Related | 898 | 242 | 26.9 | 24.1 | 30.0 | 299 | 89 | 29.8 | 24.6 | 35.3 |
| Diarrhoea | All | 898 | 22 | 2.4 | 1.5 | 3.7 | 299 | 8 | 2.7 | 1.2 | 5.2 |
| | Grade 3 | 898 | 5 | 0.6 | 0.2 | 1.3 | 299 | 3 | 1.0 | 0.2 | 2.9 |
| | Related | 898 | 22 | 2.4 | 1.5 | 3.7 | 299 | 8 | 2.7 | 1.2 | 5.2 |
| Fever(°C) | All | 898 | 253 | 28.2 | 25.3 | 31.2 | 299 | 74 | 24.7 | 20.0 | 30.0 |
| ` ' | Grade 3 | 898 | 4 | 0.4 | 0.1 | 1.1 | 299 | 3 | 1.0 | 0.2 | 2.9 |
| | Related | 898 | 246 | 27.4 | 24.5 | 30.4 | 299 | 71 | 23.7 | 19.0 | 29.0 |
| Irritability | All | 898 | 627 | 69.8 | 66.7 | 72.8 | 299 | 200 | 66.9 | 61.2 | 72.2 |
| • | Grade 3 | 898 | 43 | 4.8 | 3.5 | 6.4 | 299 | 12 | 4.0 | 2.1 | 6.9 |
| | Related | 898 | 615 | 68.5 | 65.3 | 71.5 | 299 | 196 | 65.6 | 59.9 | 70.9 |
| Loss of appetite | All | 898 | 202 | 22.5 | 19.8 | 25.4 | 299 | 62 | 20.7 | 16.3 | 25.8 |
| | Grade 3 | 898 | 1 | 0.1 | 0.0 | 0.6 | 299 | 0 | 0.0 | 0.0 | 1.2 |
| | Related | 898 | 194 | 21.6 | 19.0 | 24.4 | 299 | 60 | 20.1 | 15.7 | 25.1 |
| Vomiting | All | 898 | 116 | 12.9 | 10.8 | 15.3 | 299 | 41 | 13.7 | 10.0 | 18.1 |
| | Grade 3 | 898 | 23 | 2.6 | 1.6 | 3.8 | 299 | 11 | 3.7 | 1.9 | 6.5 |
| | Related | 898 | 112 | 12.5 | 10.4 | 14.8 | 299 | 40 | 13.4 | 9.7 | 17.8 |

LIQPOOL = Pooled HRV vaccine liquid formulation

HRV LYO = HRV vaccine HRV Lyophilised formulation

N = number of subjects having received the considered dose

n/% = number/percentage of subjects reporting the specified symptom for the considered dose

All = any occurrence of the specified symptom, irrespective of intensity grade and relationship to vaccination

Grade 3 = any occurrence of the specified symptom rated as grade 3

Related = any occurrence of the specified symptom assessed as causally related to the vaccination

95% CI = Exact 95% Confidence Interval; LL = Lower Limit, UL = Upper Limit

116194 [DTPA-IPV (INFANRIX-IPV)-061] Statistical Analysis Plan Amendment 2 Final

Template 15 Percentage of subjects reporting each solicited general symptom including those rated grade 3 in intensity and those assessed as related to vaccination during the 8-day (Day 0 to Day 7) follow-up period, for each dose in the pooled HRV vaccine liquid formulation group and the HRV vaccine HRV Lyophilised formulation group - TVC

| | | | | LIQPO | OL | | | | HRV L | <b>/</b> 0 | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | | | 95 9 | % CI | | | | 95 9 | % CI |
| Symptom | Туре | N | n | % | LL | UL | N | n | % | LL | UL |
| | | | ٥v | erall/do | se | | | | | | |
| Cough/runny nose | All | 900 | 233 | 25.9 | 23.1 | 28.9 | 300 | 79 | 26.3 | 21.4 | 31.7 |
| | Grade 3 | 900 | 2 | 0.2 | 0.0 | 0.8 | 300 | 4 | 1.3 | 0.4 | 3.4 |
| | Related | 900 | 187 | 20.8 | 18.2 | 23.6 | 300 | 64 | 21.3 | 16.8 | 26.4 |
| Diarrhoea | All | 900 | 25 | 2.8 | 1.8 | 4.1 | 300 | 4 | 1.3 | 0.4 | 3.4 |
| | Grade 3 | 900 | 7 | 8.0 | 0.3 | 1.6 | 300 | 1 | 0.3 | 0.0 | 1.8 |
| | Related | 900 | 25 | 2.8 | 1.8 | 4.1 | 300 | 3 | 1.0 | 0.2 | 2.9 |
| Fever(°C) | All | 900 | 179 | 19.9 | 17.3 | 22.6 | 300 | 68 | 22.7 | 18.1 | 27.8 |
| | Grade 3 | 900 | 2 | 0.2 | 0.0 | 0.8 | 300 | 0 | 0.0 | 0.0 | 1.2 |
| | Related | 900 | 174 | 19.3 | 16.8 | 22.1 | 300 | 67 | 22.3 | 17.7 | 27.5 |
| Irritability | All | 900 | 629 | 69.9 | 66.8 | 72.9 | 300 | 207 | 69.0 | 63.4 | 74.2 |
| | Grade 3 | 900 | 38 | 4.2 | 3.0 | 5.7 | 300 | 12 | 4.0 | 2.1 | 6.9 |
| | Related | 900 | 607 | 67.4 | 64.3 | 70.5 | 300 | 201 | 67.0 | 61.4 | 72.3 |
| Loss of appetite | All | 900 | 231 | 25.7 | 22.8 | 28.7 | 300 | 67 | 22.3 | 17.7 | 27.5 |
| | Grade 3 | 900 | 1 | 0.1 | 0.0 | 0.6 | 300 | 1 | 0.3 | 0.0 | 1.8 |
| | Related | 900 | 220 | 24.4 | 21.7 | 27.4 | 300 | 63 | 21.0 | 16.5 | 26.1 |
| Vomiting | All | 900 | 136 | 15.1 | 12.8 | 17.6 | 300 | 55 | 18.3 | 14.1 | 23.2 |
| | Grade 3 | 900 | 25 | 2.8 | 1.8 | 4.1 | 300 | 11 | 3.7 | 1.8 | 6.5 |
| | Related | 900 | 127 | 14.1 | 11.9 | 16.6 | 300 | 51 | 17.0 | 12.9 | 21.7 |

LIQPOOL = Pooled HRV vaccine liquid formulation

HRV LYO = HRV vaccine HRV Lyophilised formulation

N = number of subjects having received the considered dose

n/% = number/percentage of subjects reporting the specified symptom for the considered dose

All = any occurrence of the specified symptom, irrespective of intensity grade and relationship to vaccination

Grade 3 = any occurrence of the specified symptom rated as grade 3

Related = any occurrence of the specified symptom assessed as causally related to the vaccination

95% CI = Exact 95% Confidence Interval; LL = Lower Limit, UL = Upper Limit

116194 [DTPA-IPV (INFANRIX-IPV)-061] Statistical Analysis Plan Amendment 2 Final

Template 16 Incidence of any large injection site reaction (defined as a swelling with a diameter > 100 mm, noticeable diffuse swelling or noticeable increase in limb circumference) with onset within 4 days (Day 0–3) after booster vaccination (Total Vaccinated Cohort at Year 9)

| | (Eac | h group)<br>N= | | | | Total<br>N= | |
|---|---|---|---|---|---|---|---|
| n | % | 95%CI | | n | % | 95% CI | |
| | | LL | UL | | | LL | UL |
| | n | | | N=<br>n % 95%Cl | N=<br>n % 95%Cl n | N= | N= N= n % 95%CI n % 95% CI |

Boostrix group= Subjects who had received GSK Biologicals' Tdap vaccine (Boostrix) in study 106316 and a second dose of Tdap vaccine (Boostrix) at Year 9 Visit 6

Adacel group= Subjects who had received Sanofi Pasteurs' Tdap vaccine (Adacel) in study 106316 and a second dose of Tdap vaccine (Boostrix) at Year 9 Visit 6

Control group= Subjects who will receive the first dose of Tdap vaccine (Boostrix) at Year 9 Visit 6

N = Number of subjects with documented dose

n/% = number/percentage of subjects reporting a specified symptom

95% CI = Exact 95% confidence interval, LL = Lower Limit, UL = Upper Limit

116194 [DTPA-IPV (INFANRIX-IPV)-061] Statistical Analysis Plan Amendment 2 Final

Template 17 Percentage of subjects with grade 3 unsolicited symptoms classified by MedDRA SOC and PT from Day 0 to Day 30 after any vaccination in each HRV vaccine liquid formulation group - TVC

| | | HRV<br>N = | - | | | | V LIQ<br>= 302 | | | | V LIQ<br>= 300 | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | | 95% | CI | | | 95% | CI | | | 95% | CI |
| Primary System Organ<br>Class (CODE) | Preferred<br>Term (CODE) | n | % | LL | UL | n | % | LL | UL | n | % | LL | UL |
| At least one symptom | , | 24 | 8.1 | 5.2 | 11.7 | 26 | 8.6 | 5.7 | 12.4 | 33 | 11.0 | 7.7 | 15.1 |
| Ear and labyrinth disorders (10013993) | Ear pain<br>(10014020) | 0 | 0.0 | 0.0 | 1.2 | 1 | 0.3 | 0.0 | 1.8 | 0 | 0.0 | 0.0 | 1.2 |
| Eye disorders<br>(10015919) | Conjunctivitis (10010741) | 1 | 0.3 | 0.0 | 1.9 | 1 | 0.3 | 0.0 | 1.8 | 1 | 0.3 | 0.0 | 1.8 |
| Gastrointestinal disorders (10017947) | Diarrhoea (10012735) | 0 | 0.0 | 0.0 | 1.2 | 2 | 0.7 | 0.1 | 2.4 | 1 | 0.3 | 0.0 | 1.8 |
| a.co. a.c. (100110111) | Flatulence (10016766) | 1 | 0.3 | 0.0 | 1.9 | 1 | 0.3 | 0.0 | 1.8 | 2 | 0.7 | 0.1 | 2.4 |
| General disorders and administration site conditions (10018065) | Injection site erythema (10022061) | 0 | 0.0 | 0.0 | 1.2 | 0 | 0.0 | 0.0 | 1.2 | 1 | 0.3 | 0.0 | 1.8 |
| | Injection site pain (10022086) | 0 | 0.0 | 0.0 | 1.2 | 0 | 0.0 | 0.0 | 1.2 | 1 | 0.3 | 0.0 | 1.8 |
| | Injection site<br>swelling<br>(10053425) | 0 | 0.0 | 0.0 | 1.2 | 0 | 0.0 | 0.0 | 1.2 | 1 | 0.3 | 0.0 | 1.8 |
| | Irritability<br>(10022998) | 0 | 0.0 | 0.0 | 1.2 | 1 | 0.3 | 0.0 | 1.8 | 1 | 0.3 | 0.0 | 1.8 |
| | Pyrexia (10037660) | 4 | 1.3 | 0.4 | 3.4 | 3 | 1.0 | 0.2 | 2.9 | 4 | 1.3 | 0.4 | 3.4 |
| Immune system disorders (10021428) | Hypersensitivity (10020751) | 0 | 0.0 | 0.0 | 1.2 | 1 | 0.3 | 0.0 | 1.8 | 0 | 0.0 | 0.0 | 1.2 |
| Infections and infestations (10021881) | Bronchitis<br>(10006451) | 2 | 0.7 | 0.1 | 2.4 | 0 | 0.0 | 0.0 | 1.2 | 1 | 0.3 | 0.0 | 1.8 |
| | Ear infection (10014011) | 1 | 0.3 | 0.0 | 1.9 | 3 | 1.0 | 0.2 | 2.9 | 2 | 0.7 | 0.1 | 2.4 |
| | Exanthema<br>subitum<br>(10015586) | 1 | 0.3 | 0.0 | 1.9 | 1 | 0.3 | 0.0 | 1.8 | 0 | 0.0 | 0.0 | 1.2 |
| | Eye infection (10015929) | 1 | 0.3 | 0.0 | 1.9 | 0 | 0.0 | 0.0 | 1.2 | 0 | 0.0 | 0.0 | 1.2 |
| | Gastroenteritis (10017888) | 0 | 0.0 | 0.0 | 1.2 | 0 | 0.0 | 0.0 | 1.2 | 1 | 0.3 | 0.0 | 1.8 |
| | Impetigo<br>(10021531) | 1 | 0.3 | 0.0 | 1.9 | 0 | 0.0 | 0.0 | 1.2 | 0 | 0.0 | 0.0 | 1.2 |
| | Influenza<br>(10022000) | 0 | 0.0 | 0.0 | 1.2 | 1 | 0.3 | 0.0 | 1.8 | 0 | 0.0 | 0.0 | 1.2 |
| | Laryngitis<br>(10023874) | 1 | 0.3 | 0.0 | 1.9 | 0 | 0.0 | 0.0 | 1.2 | 0 | 0.0 | 0.0 | 1.2 |
| | Otitis media (10033078) | 5 | 1.7 | 0.5 | 3.9 | 6 | 2.0 | | 4.3 | 11 | 3.7 | 1.8 | 6.5 |
| | Perianal<br>abscess<br>(10034447) | 1 | 0.3 | 0.0 | 1.9 | 0 | 0.0 | 0.0 | 1.2 | 0 | 0.0 | 0.0 | 1.2 |
| | Pneumonia<br>(10035664) | 0 | 0.0 | 0.0 | 1.2 | 1 | 0.3 | 0.0 | 1.8 | 0 | 0.0 | 0.0 | 1.2 |

116194 [DTPA-IPV (INFANRIX-IPV)-061] Statistical Analysis Plan Amendment 2 Final

| | | | | | Stati | istica | al Ana | ilysis | Plan | Am | endm | ent 2 | Final |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | HRV | 'LIQ | | | HR | V LIQ | | | HR | V LIQ | | |
| | | N = | 298 | | | N: | = 302 | | | N: | = 300 | | |
| | | | | 95% | CI | | | 95% | CI | | | 95% | CI |
| Primary System Organ | Preferred | n | % | LL | UL | n | % | LL | UL | n | % | LL | UL |
| Class (CODE) | Term (CODE) | | | | | | | | | | | | |
| | Respiratory | 3 | 1.0 | 0.2 | 2.9 | 2 | 0.7 | 0.1 | 2.4 | 0 | 0.0 | 0.0 | 1.2 |
| | tract infection | | | | | | | | | | | | |
| | (10062352) | | | | | | | | | | | | |
| | Respiratory | 0 | 0.0 | 0.0 | 1.2 | 0 | 0.0 | 0.0 | 1.2 | 1 | 0.3 | 0.0 | 1.8 |
| | tract infection | | | | | | | | | | | | |
| | viral | | | | | | | | | | | | |
| | (10062106) | | | | | | | | | | | | |
| | Rhinitis | 2 | 0.7 | 0.1 | 2.4 | 1 | 0.3 | 0.0 | 1.8 | 3 | 1.0 | 0.2 | 2.9 |
| | (10039083) | | | | | | | | | | | | |
| | Upper | 2 | 0.7 | 0.1 | 2.4 | 5 | 1.7 | 0.5 | 3.8 | 7 | 2.3 | 0.9 | 4.7 |
| | respiratory tract | | | | | | | | | | | | |
| | infection | | | | | | | | | | | | |
| | (10046306) | | | | | | | | | | | | |
| | Varicella | 0 | 0.0 | 0.0 | 1.2 | 1 | 0.3 | 0.0 | 1.8 | 2 | 0.7 | 0.1 | 2.4 |
| | (10046980) | | | | | | | | | | | | |
| Psychiatric disorders | Crying | 0 | 0.0 | 0.0 | 1.2 | 0 | 0.0 | 0.0 | 1.2 | 1 | 0.3 | 0.0 | 1.8 |
| (10037175) | (10011469) | | 0.0 | | 4.0 | | 0.0 | | 4.0 | _ | 0.0 | | 4.0 |
| Respiratory, thoracic | Cough | 1 | 0.3 | 0.0 | 1.9 | 1 | 0.3 | 0.0 | 1.8 | 6 | 2.0 | 0.7 | 4.3 |
| and mediastinal | (10011224) | | | | | | | | | | | | |
| disorders (10038738) | N | | 0.0 | 0.0 | 4.0 | _ | 0.0 | 0.0 | 4.0 | _ | 0.0 | 0.0 | 4.0 |
| | Nasal | 1 | 0.3 | 0.0 | 1.9 | 0 | 0.0 | 0.0 | 1.2 | 0 | 0.0 | 0.0 | 1.2 |
| | congestion | | | | | | | | | | | | |
| | (10028735) | 0 | 0.0 | 0.0 | 1.2 | 0 | 0.0 | 0.0 | 1.2 | 1 | 0.3 | 0.0 | 1.8 |
| | Rales | U | 0.0 | 0.0 | 1.2 | U | 0.0 | 0.0 | 1.2 | 1 | 0.3 | 0.0 | 1.0 |
| Skin and subcutaneous | (10037833) | 1 | 0.3 | 0.0 | 1.9 | 1 | 0.3 | 0.0 | 1.8 | 0 | 0.0 | 0.0 | 1.2 |
| tissue disorders | Dermatitis | 1 | 0.3 | 0.0 | 1.9 | | 0.3 | 0.0 | 1.0 | U | 0.0 | 0.0 | 1.2 |
| (10040785) | allergic<br>(10012434) | | | | | | | | | | | | |
| (10040703) | Eczema | 0 | 0.0 | 0.0 | 1.2 | 0 | 0.0 | 0.0 | 1.2 | 1 | 0.3 | 0.0 | 1.8 |
| | (10014184) | U | 0.0 | 0.0 | 1.2 | U | 0.0 | 0.0 | 1.2 | 1 | 0.5 | 0.0 | 1.0 |
| | Rash | 2 | 0.7 | 0.1 | 2.4 | 0 | 0.0 | 0.0 | 1.2 | 0 | 0.0 | 0.0 | 1.2 |
| | (10037844) | _ | 0.1 | 0.1 | 2.4 | U | 0.0 | 0.0 | 1.2 | U | 0.0 | 0.0 | 1.2 |
| | (10001044) | l | | | | | | | 1 | | | | |

HRV LIQ = HRV vaccine liquid formulation Lot A

HRV LIQ = HRV vaccine liquid formulation Lot B HRV LIQ = HRV vaccine liquid formulation Lot C

N = number of subjects with at least one administered dose

n/% = number/percentage of subjects reporting at least once a specified unsolicited symptom
At least one symptom = number of subjects reporting at least one unsolicited symptom, whatever the MedDRA PT
95% CI = exact 95% Confidence Interval, LL = Lower Limit, UL = Upper Limit

116194 [DTPA-IPV (INFANRIX-IPV)-061] Statistical Analysis Plan Amendment 2 Final

Template 18 Percentage of doses with grade 3 unsolicited symptoms classified by MedDRA SOC and PT from Day 0 to Day 30 after vaccination in each HRV vaccine liquid formulation group - TVC

| | | | | V LIQ<br>= 603 | | | | / LIQ<br>: 600 | |
|---|---|---|---|---|---|---|---|---|---|
| | | | | 959 | % CI | | | 959 | % CI |
| Primary System Organ<br>Class (CODE) | Preferred Term (CODE) | n | % | LL | UL | n | % | LL | UL |
| At least one symptom | | 30 | 5.0 | 3.4 | 7.0 | 38 | 6.3 | 4.5 | 8.6 |
| Ear and labyrinth<br>disorders (10013993) | Ear pain (10014020) | 1 | 0.2 | 0.0 | 0.9 | 0 | 0.0 | 0.0 | 0.6 |
| Eye disorders (10015919) | Conjunctivitis (10010741) | 1 | 0.2 | 0.0 | 0.9 | 1 | 0.2 | 0.0 | 0.9 |
| Gastrointestinal disorders (10017947) | Diarrhoea (10012735) | 2 | 0.3 | 0.0 | 1.2 | 1 | 0.2 | 0.0 | 0.9 |
| | Flatulence (10016766) | 1 | 0.2 | 0.0 | 0.9 | 2 | 0.3 | 0.0 | 1.2 |
| General disorders and administration site conditions (10018065) | Injection site erythema (10022061) | 0 | 0.0 | 0.0 | 0.6 | 1 | 0.2 | 0.0 | 0.9 |
| , | Injection site pain (10022086) | 0 | 0.0 | 0.0 | 0.6 | 1 | 0.2 | 0.0 | 0.9 |
| | Injection site swelling (10053425) | 0 | 0.0 | 0.0 | 0.6 | 1 | 0.2 | 0.0 | 0.9 |
| | Irritability (10022998) | 1 | 0.2 | 0.0 | 0.9 | 1 | 0.2 | 0.0 | 0.9 |
| | Pyrexia (10037660) | 3 | 0.5 | 0.1 | 1.4 | 4 | 0.7 | 0.2 | 1.7 |
| Immune system disorders (10021428) | Hypersensitivity (10020751) | 1 | 0.2 | 0.0 | 0.9 | 0 | 0.0 | 0.0 | 0.6 |
| Infections and infestations (10021881) | Bronchitis (10006451) | 0 | 0.0 | 0.0 | 0.6 | 1 | 0.2 | 0.0 | 0.9 |
| , | Ear infection (10014011) | 3 | 0.5 | 0.1 | 1.4 | 2 | 0.3 | 0.0 | 1.2 |
| | Exanthema subitum (10015586) | 1 | 0.2 | 0.0 | 0.9 | 0 | 0.0 | 0.0 | 0.6 |
| | Eye infection (10015929) | 0 | 0.0 | 0.0 | 0.6 | 0 | 0.0 | 0.0 | 0.6 |
| | Gastroenteritis (10017888) | 0 | 0.0 | 0.0 | 0.6 | 1 | 0.2 | 0.0 | 0.9 |
| | Impetigo (10021531) | 0 | 0.0 | 0.0 | 0.6 | 0 | 0.0 | 0.0 | 0.6 |
| | Influenza (10022000) | 1 | 0.2 | 0.0 | 0.9 | 0 | 0.0 | 0.0 | 0.6 |
| | Laryngitis (10023874) | 0 | 0.0 | 0.0 | 0.6 | 0 | 0.0 | 0.0 | 0.6 |
| | Otitis media (10033078) | 7 | 1.2 | 0.5 | 2.4 | 12 | 2.0 | 1.0 | 3.5 |
| | Perianal abscess (10034447) | 0 | 0.0 | 0.0 | 0.6 | 0 | 0.0 | 0.0 | 0.6 |
| | Pneumonia (10035664) | 1 | 0.2 | 0.0 | 0.9 | 0 | 0.0 | 0.0 | 0.6 |
| | Respiratory tract infection (10062352) | 2 | 0.3 | 0.0 | 1.2 | 0 | 0.0 | 0.0 | 0.6 |
| | Respiratory tract infection viral (10062106) | 0 | 0.0 | 0.0 | 0.6 | 1 | 0.2 | 0.0 | 0.9 |
| | Rhinitis (10039083) | 1 | 0.2 | 0.0 | 0.9 | 3 | 0.5 | 0.1 | 1.5 |
| | Upper respiratory tract infection (10046306) | 6 | 1.0 | 0.4 | 2.2 | 8 | 1.3 | 0.6 | 2.6 |
| | Varicella (10046980) | 1 | 0.2 | 0.0 | 0.9 | 2 | 0.3 | 0.0 | 1.2 |
| Psychiatric disorders<br>(10037175) | Crying (10011469) | 0 | 0.0 | 0.0 | 0.6 | 1 | 0.2 | 0.0 | 0.9 |
| Respiratory, thoracic and mediastinal disorders | Cough (10011224) | 1 | 0.2 | 0.0 | 0.9 | 6 | 1.0 | 0.4 | 2.2 |
| (10038738) | Nasal congestion (10028735) | 0 | 0.0 | 0.0 | 0.6 | 0 | 0.0 | 0.0 | 0.6 |
| . , | Rales (10037833) | 0 | 0.0 | 0.0 | 0.6 | 1 | 0.2 | 0.0 | 0.9 |
| Skin and subcutaneous tissue disorders | Dermatitis allergić (10012434) | 1 | 0.2 | 0.0 | 0.9 | 0 | 0.0 | 0.0 | 0.6 |

116194 [DTPA-IPV (INFANRIX-IPV)-061] Statistical Analysis Plan Amendment 2 Final

| | | | | V LIQ<br>= 603 | | | | / LIQ<br>: 600 | |
|---|---|---|---|---|---|---|---|---|---|
| | | | | 95 | % CI | | | 95 | % CI |
| Primary System Organ<br>Class (CODE) | Preferred Term (CODE) | n | % | LL | UL | n | % | LL | UL |
| (10040785) | Eczema (10014184) | 0 | 0.0 | 0.0 | 0.6 | 1 | 0.2 | 0.0 | 0.9 |
| | Rash (10037844) | 0 | 0.0 | 0.0 | 0.6 | 0 | 0.0 | 0.0 | 0.6 |

HRV LIQ = HRV vaccine liquid formulation Lot A

HRV LIQ = HRV vaccine liquid formulation Lot B

HRV LIQ = HRV vaccine liquid formulation Lot C

N = Total number of doses administered

n/% = number/percentage of doses followed by at least one report of the specified unsolicited symptom
At least one symptom = number of doses followed by at least one report of an unsolicited symptom whatever the
MedDRA PT

95% CI = Exact 95% Confidence Interval; LL = Lower Limit, UL = Upper Limit

Template 19 Number (%) of subjects with serious adverse events from first study vaccination up to Visit 3 including number of events reported (TVC)

| | | | | Gr<br>N = | - | | Gr.<br>N | _ |
|---|---|---|---|---|---|---|---|---|
| Type of Event | Primary System Organ<br>Class | Preferred Term<br>(CODE) | n* | n | % | n* | n | % |
| SAE | At least one symptom | | | | | | | |
| | <each soc=""></each> | <each pt="" term=""></each> | | | | | | |
| Related SAE | At least one symptom | | | | | | | |
| | <each soc=""></each> | <each pt="" term=""></each> | | | | | | |
| Fatal SAE | At least one symptom | | | | | | | |
| | <each soc=""></each> | <each pt="" term=""></each> | | | | | | |
| Related fatal SAE | At least one symptom | | | | | | | |
| | <each soc=""></each> | <each pt="" term=""></each> | | | | | | |

Gr 1 = Group 1 description

Gr 2 = Group 2 description

N = number of subjects with the administered dose

n\* = number of events reported

n/% = number/percentage of subjects reporting the symptom at least once

116194 [DTPA-IPV (INFANRIX-IPV)-061] Statistical Analysis Plan Amendment 2 Final

# Template 20 Subjects with Serious Adverse Events reported up to Visit 3 - TVC

| Sub.<br>No. | Case Id | Age at onset (Week) | Sex | Verbatim | Preferred term | System Organ<br>Class | MA<br>type | Dose | Day of onset | Duration | Causality | Outcome |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| P<br>P | PPD | 12 | М | Kawasaki's<br>disease | Kawasaki's<br>disease | Infections and infestations | НО | 1 | 12 | 29 | N | Recovered/resolved |
| PP<br>D | PPD | 18 | M | Influenza-b | Influenza | Infections and infestations | НО | 2 | 2 | 5 | N | Recovered/resolved |
| PP<br>D | PPD | 17 | M | Acute gastroenteritis | Gastroenteritis | Infections and infestations | НО | 2 | 9 | 5 | N | Recovered/resolved |
| PP<br>D | PPD | 17 | F | Infantile spasms | Infantile spasms | Nervous system disorders | НО | 2 | 2 | 51 | N | Recovered/resolved with sequelae |
| PP<br>D | PPD | 21 | М | | Respiratory syncytial virus bronchiolitis | Infections and infestations | НО | 2 | 30 | 16 | N | Recovered/resolved |
| PP<br>D | PPD | 13 | М | Gastroenteritis | Gastroenteritis | Infections and infestations | НО | 1 | 25 | 6 | N | Recovered/resolved |
| PP<br>D | PPD | 22 | М | Pneumonia | Pneumonia | Infections and infestations | НО | 2 | 32 | 13 | N | Recovered/resolved |
| | | 23 | | Middle ear infection | Otitis media | Infections and infestations | НО | 2 | 37 | 8 | N | Recovered/resolved |
| PP<br>D | PPD | 14 | F | Secretory otitis media | Otitis media | Infections and infestations | НО | 1 | 7 | 25 | N | Recovered/resolved |
| PPD | PPD | 20 | М | Viral pneumonia | Pneumonia viral | Infections and infestations | НО | 2 | 13 | 23 | N | Recovered/resolved |
| PPD | PPD | 14 | М | Middle ear infection, left | Otitis media | Infections and infestations | НО | 1 | 19 | 8 | N | Recovered/resolved |
| | | 14 | | Pneumonia | Pneumonia | Infections and infestations | НО | 1 | 19 | 8 | N | Recovered/resolved |
| PPD | PPD | 13 | М | Acute lymphadenitis | Lymphadenitis | Blood and lymphatic system disorders | НО | 1 | 13 | 22 | N | Recovered/resolved |
| PPD | PPD | 10 | F | Pyelonephritis | Pyelonephritis acute | Infections and infestations | НО | 1 | 6 | 12 | N | Recovered/resolved |
| PPD | PPD | 19 | М | Laryngitis | Laryngitis | Infections and infestations | НО | 2 | 11 | 7 | N | Recovered/resolved |
| PPD | PPD | 14 | M | Bronchitis acuta | Bronchitis | Infections and | НО | 1 | 23 | 12 | N | Recovered/resolved |

# 116194 [DTPA-IPV (INFANRIX-IPV)-061] Statistical Analysis Plan Amendment 2 Final

| Sub.<br>No. | Case Id | Age at onset (Week) | | Verbatim | Preferred term | System Organ<br>Class | MA<br>type | Dose | Day of onset | Duration | Causality | Outcome |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | | | | infestations | | | | | | |
| PPD | PPD | 19 | М | Bronchiolitis acuta | Bronchiolitis | Infections and infestations | НО | 2 | 26 | 7 | N | Recovered/resolved |
| PPD | PPD | 19 | F | Laryngitis acuta | Laryngitis | Infections and infestations | НО | 2 | 7 | 4 | N | Recovered/resolved |
| PPD | PPD | 18 | F | Laryngitis | Laryngitis | Infections and infestations | НО | 2 | 7 | 4 | N | Recovered/resolved |
| PPD | PPD | 14 | F | Gastroenteritis | Gastroenteritis | Infections and infestations | НО | 1 | 22 | 7 | N | Recovered/resolved |

MA = medical attention

HO = hospitalisation

Dose = dose given prior to the start of the SAE

Day of onset = number of days since last study vaccine dose

14-DEC-2017 Page 48 of 51

116194 [DTPA-IPV (INFANRIX-IPV)-061] Statistical Analysis Plan Amendment 2 Final

Template 21 Number and percentage of doses and of subjects who took at least one concomitant medication from Day 0 to Day 7 after vaccination by type in each HRV vaccine liquid formulation group - TVC

| | HRV LIQ | | | | | HRV LIQ | | | | HRV LIQ | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | | 95% | 6 CI | | | | 95% | 6 CI | | | | 95% CI | |
| | N | n | % | LL | UL | N | n | % | LL | UL | N | n | % | LL | UL |
| Dose 1 | | | | | | | | | | | | | | | |
| Any | 298 | 173 | 58.1 | 52.2 | 63.7 | 302 | 175 | 57.9 | 52.2 | 63.6 | 300 | 157 | 52.3 | 46.5 | 58.1 |
| Any antipyretic | 298 | 97 | 32.6 | 27.3 | 38.2 | 302 | 94 | 31.1 | 25.9 | 36.7 | 300 | 71 | 23.7 | 19.0 | 28.9 |
| Prophylactic antipyretic | 298 | 8 | 2.7 | 1.2 | 5.2 | 302 | 6 | 2.0 | 0.7 | 4.3 | 300 | 9 | 3.0 | 1.4 | 5.6 |
| Dose 2 | | | | | | | | | | | | | | | |
| Any | 297 | 105 | 35.4 | 29.9 | 41.1 | 301 | 117 | 38.9 | 33.3 | 44.6 | 300 | 89 | 29.7 | 24.6 | 35.2 |
| Any antipyretic | 297 | 98 | 33.0 | 27.7 | 38.7 | 301 | 109 | 36.2 | 30.8 | 41.9 | 300 | 86 | 28.7 | 23.6 | 34.1 |
| Prophylactic | 297 | 7 | 2.4 | 1.0 | 4.8 | 301 | 8 | 2.7 | 1.2 | 5.2 | 300 | 6 | 2.0 | 0.7 | 4.3 |
| antipyretic | | | | | | | | | | | | | | | |
| | | | | | ( | Overa | III/do: | se | | | | | | | |
| Any | 595 | 278 | 46.7 | 42.7 | 50.8 | 603 | 292 | 48.4 | 44.4 | 52.5 | 600 | 246 | 41.0 | 37.0 | 45.1 |
| Any antipyretic | 595 | 195 | 32.8 | 29.0 | 36.7 | 603 | 203 | 33.7 | 29.9 | 37.6 | 600 | 157 | 26.2 | 22.7 | 29.9 |
| Prophylactic | 595 | 15 | 2.5 | 1.4 | 4.1 | 603 | 14 | 2.3 | 1.3 | 3.9 | 600 | 15 | 2.5 | 1.4 | 4.1 |
| antipyretic | | | | | | | | | | | | | | | |
| | | | | | 0 | veral | l/subj | ject | | | | | | | |
| Any | 298 | 194 | 65.1 | 59.4 | 70.5 | 302 | 205 | 67.9 | 62.3 | 73.1 | 300 | 182 | 60.7 | 54.9 | 66.2 |
| Any antipyretic | 298 | 130 | 43.6 | 37.9 | 49.5 | 302 | 141 | 46.7 | 41.0 | 52.5 | 300 | 111 | 37.0 | 31.5 | 42.7 |
| Prophylactic | 298 | 11 | 3.7 | 1.9 | 6.5 | 302 | 12 | 4.0 | 2.1 | 6.8 | 300 | 13 | 4.3 | 2.3 | 7.3 |
| antipyretic | | | | | | | | | | | | | | | |

HRV LIQ = HRV vaccine liquid formulation Lot A

HRV LIQ = HRV vaccine liquid formulation Lot B

HRV LIQ = HRV vaccine liquid formulation Lot C

For each dose and overall/subject:

N = number of subjects with at least one administered dose

n/% = number/percentage of subjects who started to take the specified concomitant medication at least once during the mentioned period

For overall/dose:

N = number of administered doses

n/% = number/percentage of doses after which the specified concomitant medication was started at least once during the mentioned period

95% CI = exact 95% Confidence Interval, LL = Lower Limit, UL = Upper Limit

116194 [DTPA-IPV (INFANRIX-IPV)-061] Statistical Analysis Plan Amendment 2 Final

Template 22 Solicited and Unsolicited symptoms experienced by at least 5 % of subjects classified by MedDRA Primary System Organ Class and Preferred Term within the 31-day (Days 0-30) post-vaccination period - AE below 5 % and SAE excluded (Total vaccinated cohort)

| | | | HPV<br>N | | MN | IR_D<br>N = | |
|---|---|---|---|---|---|---|---|
| Primary System Organ Class (CODE) | Preferred Term (CODE) | n* | n | % | n* | n | % |
| At least one symptom | | | | | | | |
| <each soc=""></each> | <each pt="" term=""></each> | | | | | | |

HPV\_2D = females aged 4-6 years who received two doses of HPV-16/18 L1 VLP AS04 vaccine at Day 0 and Month 6 MMR\_DTPa = females aged 4-6 years who received MMR vaccine at Day 0 and DTPa vaccine at Month 6

At least one symptom = at least one symptom experienced (regardless of the MedDRA Preferred Term)

N = number of subjects with the administered dose

n\* = number of events reported

n/% = number/percentage of subjects reporting the symptom at least once

95% CI = exact 95% confidence interval; LL = Lower Limit, UL = Upper Limit

### Template 23 Minimum and maximum activity dates (TVC)

| Visit | Minimum date | Maximum date |
|-------|--------------|--------------|
| 1 | 19JUN2007 | 29DEC2007 |
| 2 | 24JUL2007 | 08FEB2008 |
| 3 | 24AUG2007 | 18MAR2008 |
| 4 | 25MAR2008 | 22NOV2008 |
| 5 | 24MAR2009 | 31MAR2009* |

<sup>\*</sup>Database Lock Date = 31MAR2009

# Template 24 Number of enrolled subjects by age category (TVC)

| | | Gr 1<br>N = | Gr 2<br>N = | Gr 3<br>N = | Total<br>N = |
|---|---|---|---|---|---|
| Characteristics | Categories | n | n | n | n |
| Age category | In utero | | | | |
| | Preterm newborn infants | | | | |
| | (gestational age < 37 wks) | | | | |
| | Newborns (0-27 days) | | | | |
| | Infants and toddlers (28 days-23 months) | | | | |
| | Children (2-11 years) | | | | |
| | Adolescents (12-17 years) | | | | |
| | Adults (18-64 years) | | | | |
| | From 65-84 years | | | | |
| | 85 years and over | | | | |
| | Missing | | | | |

Gr 1 = Group 1 description

Gr 2 = Group 2 description

Gr 3 = Group 3 description

N = Number of enrolled subjects

n= number of enrolled subjects included in each group or in total for a given age category or for all age categories Missing = <describe missing>

116194 [DTPA-IPV (INFANRIX-IPV)-061] Statistical Analysis Plan Amendment 2 Final

# Template 25 Number of subjects by country

| | ACWY-TT<br>N = 259 | ACWYHPV<br>N = 259 | HPV<br>N = 261 | Co-ad<br>N = 260 | Tdap<br>N = 261 | Total<br>N = 1300 |
|---|---|---|---|---|---|---|
| Country | n | n | N | n | n | n |
| Dominican Republic | 86 | 87 | 88 | 87 | 87 | 435 |
| Estonia | 87 | 86 | 87 | 87 | 88 | 435 |
| Thailand | 86 | 86 | 86 | 86 | 86 | 430 |

ACWY-TT = Subjects who received MenACWY-TT at Month 0 and Cervarix at Month 1, 2 and 7

ACWYHPV = Subjects who received MenACWY-TT and Cervarix at Month 0 and Cervarix at Month 1 and 6 HPV = Subjects who received Cervarix at Month 0, 1 and 6

Co-ad = Subjects who received MenACWY-TT, Cervarix and Boostrix at Month 0 and Cervarix at Month 1 and 6 Tdap = Subjects who received Boostrix and Cervarix at Month 0 and Cervarix at Month 1 and 6 N = number of subjects

n= number of enrolled subjects included in each group or in total for a given age category or for all age categories

# Template 26 Listing of dropouts due to AEs, SAEs and solicited symptoms (Total cohort)

| Study-<br>Subject | Country | Gender | AE Description | SAE | Causality | Outcome | Type of discontinuation |
|---|---|---|---|---|---|---|---|
| No.<br>PP | Germany | F | SUBJECT DIED | Υ | | | Study at visit/contact:<br>VISIT11 (Y5) |
| PP<br>D | Germany | F | SUBJECT DIED | Υ | | | Study at visit/contact:<br>VISIT11 (Y5) |